# **Statistical Analysis Plan**

Clinical trial protocol title: A phase 1, blinded, randomised, placebo-controlled,

parallel-group, single-dose, dose-escalation study to investigate safety, tolerability, and pharmacokinetics of Emodepside (BAY 44-4400) after oral dosing in healthy

male subjects

HMR code: 15-020 Part 2

Sponsor code: DNDI-EMO-001 Part 2

EudraCT no: 2015-003592-29

CRO details: Hammersmith Medicines Research

Cumberland Avenue London NW10 7EW

Sponsor details: DNDi, Chemin Louis Dunant 15, 1202 Geneva

Switzerland

Issued: 10 March 2017

Version:

Based on: Protocol version 5, Final, 18 January 2017

Number of pages: 73

Prepared by: Stephen Sah

# **Statistical Analysis Plan**

Clinical trial protocol title: A phase 1, blinded, randomised, placebo-controlled,

parallel-group, single-dose, dose-escalation study to investigate safety, tolerability, and pharmacokinetics of Emodepside (BAY 44-4400) after oral dosing in healthy

male subjects

HMR code: 15-020 Part 2

Sponsor code: DNDI-EMO-001 Part 2

EudraCT no: 2015-003592-29

CRO details: Hammersmith Medicines Research

Cumberland Avenue London NW10 7EW

Sponsor details: DNDi, Chemin Louis Dunant 15, 1202 Geneva

Switzerland

Issued: 10 March 2017

Version:

Based on: Protocol version 5, Final, 18 January 2017

Number of pages: 73

Prepared by: Stephen Sah

# **Table of contents**

| 1 | LIST | OF ABBREVIATIONS | 5 |
|----|------|------------------------------------------------------------|----|
| 2 | SIGN | NATURES | 7 |
| 3 | INTE | RODUCTION | 8 |
| 4 | STUI | DY OBJECTIVE(S) AND ENDPOINT(S) | 8 |
| | 4.1 | Study Objective(s) | |
| | | 4.1.1 Primary Objective(s) | 8 |
| | | 4.1.2 Secondary Objective(s) | 9 |
| | 4.2 | Study Endpoint(s) | 9 |
| | | 4.2.1 Safety and Tolerability Variables: | |
| | | 4.2.2 Pharmacokinetic Variables: | 10 |
| | | 4.2.3 Pharmacodynamic Variables: | |
| | 4.3 | Statistical Hypotheses | |
| 5 | STUI | DY DESIGN | 10 |
| 6 | PLA | NNED ANALYSES | 17 |
| | 6.1 | Interim Analyses | 17 |
| | | 6.1.1 Persons responsible for analysis | |
| | 6.2 | Final Analysis | 17 |
| | | 6.2.1 Persons responsible for analysis | 17 |
| 7 | SAM | PLE SIZE CONSIDERATIONS | 17 |
| | 7.1 | Sample Size Assumptions | 17 |
| 8 | ANA | LYSIS POPULATIONS | 18 |
| | 8.1 | Analysis Datasets | 18 |
| 9 | TRE | ATMENT COMPARISONS | 18 |
| | 9.1 | Data Display Treatment and Other Subgroup Descriptors | 18 |
| | | 9.1.1 Conventions for Summary Statistics and Data Displays | |
| 10 | DAT | A HANDLING CONVENTIONS | 19 |
| | 10.1 | Premature Withdrawal and Missing Data | |
| | 10.2 | Derived and Transformed Data | 20 |
| | 10.3 | Assessment Windows | 20 |
| | 10.4 | Values of Potential Clinical Importance | |
| 11 | | DY POPULATION | |
| | 11.1 | Disposition of Subjects | |
| | 11.2 | Protocol Deviations | |
| | 11.2 | Demographic and Baseline Characteristics | |
| | 11.3 | Demographic and Dascinic Characteristics | |

| | 11.4 | Treatment Compliance | 22 |
|---|---|---|---|
| 12 | SAFE | TY ANALYSES | 22 |
| | 12.1 | Extent of Exposure | 22 |
| | 12.2 | Adverse Events | 22 |
| | 12.3 | Deaths and Serious Adverse Events | 23 |
| | 12.4 | Adverse Events Leading to Withdrawal from the Study | 23 |
| | 12.5 | Clinical Laboratory Evaluations | 23 |
| | 12.6 | Other Safety Measures | 24 |
| | | 12.6.1 Vital signs | 24 |
| | | 12.6.2 ECG | 24 |
| | | 12.6.3 Neurological examination | 24 |
| | | 12.6.4 Physical examination | 24 |
| | | 12.6.5 Ophthalmology assessments | 24 |
| 13 | PHAF | RMACOKINETIC ANALYSES | 25 |
| | 13.1 | Plasma PK | 25 |
| | | 13.1.1 Pharmacokinetic Concentration Data | 25 |
| | | 13.1.2 Pharmacokinetic Parameters | 26 |
| | 13.2 | Urinary PK | 26 |
| 14 | PHAF | RMACODYNAMIC ANALYSES | 26 |
| 15 | CHAN<br>27 | NGES FROM THE PROTOCOL SPECIFIED STATISTICAL | ANALYSIS |
| 16 | REFE | CRENCES | 27 |
| 17 | ATTA | ACHMENTS | 29 |
| | 17.1 | Table of Contents for Data Display Specifications | 29 |
| | 17.2 | Data Display Specifications | |
| | -, | 17.2.1 Table Outlines | |
| | | 17.2.2 Figure Outlines | |
| | | 17.2.3 Listing Outlines | 55 |
| APPI | ENDIX | A: LABORATORY RANGES | 65 |
| APPI | ENDIX | B: PHARMACOKINETIC ANALYSIS | 67 |
| 1 | CALO | CULATION METHODS | 67 |
| | 1.1 | Data Handling Conventions | |
| | | 1.1.1 Actual v Planned Times | |
| | | 1.1.2 Missing and BQL Concentrations | |
| | 1.2 | AUC Calculations | |
| | 1.3 | Lambda-z Calculations | |
| | 1.4 | Observed v Predicted Values | |

| 2 | GEN | NERAL CONSIDERATIONS FOR DATA ANALYSIS | S69 |
|------|---------|----------------------------------------|-----|
| | 2.1 | Derived and transformed data | 69 |
| | 2.2 | Summary data | 69 |
| 3 | PAR | RAMETER DEFINITIONS | 70 |
| | 3.1 | Plasma Parameters | 70 |
| | | 3.1.1 Emodepside | 70 |
| A DI | DEMINIX | V C. SAMDI E DACE I AVOUT | 72 |



### 1 List of abbreviations

Terminal rate constant  $\lambda_z$ AΕ Adverse Event ANOVA Analysis of variance Alanine aminotransferase ALT AP Alkaline phosphatase aPTT Activated partial thromboplastin time Aspartate aminotransferase **AST AUC** Area under concentration-time curve Area under the plasma concentration-time curve from time zero to 24h  $AUC_{(0-24)}$ AUC<sub>(0-24)/D</sub> Dose-normalised AUC from time zero to 24h Area under the concentration-time curve from time zero to 24h  $AUC_{(0-24),norm}$ corrected by dose and body weight  $AUC_t$ AUC from time zero to time t  $AUC_{t-\infty}$ AUC from time t to infinity AUC from time zero (pre-dose) to the time of last quantifiable AUC<sub>t. norm</sub> concentration corrected by dose and body weight  $AUC_{\infty}$ Area under the plasma drug concentration vs. time from zero to infinity  $AUC_{\infty}/D$ The area under the plasma drug concentration vs. time curve from time zero to infinity, corrected for dose. The area under the concentration-time curve from time zero to infinity  $AUC_{\infty}$ , norm corrected by dose and body weight **BMI Body Mass Index** BP Blood pressure Below the limit of quantification **BQL** Confidence Interval CI CK Creatine kinase CL/F Apparent Total body clearance Maximum Plasma Concentration  $C_{max}$  $C_{max}/D$ C<sub>max</sub> corrected by dose C<sub>max</sub> corrected by dose and body weight  $C_{\text{max,norm}}$ Case Report Form **CRF** CTR Clinical Trial Report Coefficient of Variation CVBetween subject CV CVb ECG Electrocardiogram Glutamate dehydrogenase **GLDH** GGT Gamma-glutamyl transpeptidase HbA1C Glycated haemoglobin High-density lipoprotein **HDL** Hammersmith Medicines Research **HMR** HR Heart Rate International Conference on Harmonization **ICH** Investigational Medicinal Product **IMP** Immediate release IR Lactate dehydrogemnase LDH Low-density lipoprotein LDL Liquid Service Formulation LSF

**MCH** Hemoglobin amount per red blood cell The amount of hemoglobin relative to the size of the cell (hemoglobin **MCHC** concentration) per red blood cell **MCV** Average red blood cell size Medical Dictionary for Regulatory Activities MedDRA **MRT** Mean residence time Number of subjects N Number of observations used in analysis n PC Personal Computer Potential clinical importance **PCI** Pharmacodynamic(s) PD PK Pharmacokinetic(s) Portion of the ECG from the beginning of the P wave to the beginning PR of the QRS complex, representing atrioventricular node function. PT Prothrombin time O1 Lower quartile Q3 Upper quartile The QRS complex of the ECG reflects the rapid depolarization of the ORS right and left ventricles. QT Portion of the ECG between the onset of the Q wave and the end of the T wave, representing the total time for ventricular depolarization and repolarization. Corrected portion of the ECG between the onset of the Q wave and the QTc end of the T wave, representing the total time for ventricular depolarization and repolarization. OTc interval with Bazett's correction method **OTcB QTcF** QTc interval with Fridericia's correction method **RBC** Red blood cells RR Portion of the ECG between consecutive R waves, representing the ventricular rate Statistical Analysis Plan SAP SD Standard deviation Terminal elimination half-life  $t_{1/2}$ Dominant half-life  $t_{1/2,dom}$ TEAE Treatment-Emergent Adverse Event Time to maximum plasma concentration  $T_{max}$ Thyroid-stimulating hormone TSH Vz/FApparent volume of distribution WBC White blood cells

WHO

World Health Organisation

# 2 Signatures

The following persons have read and agreed the content of this Statistical Analysis Plan:

Stephen Sah Statistician, HMR

Malcom Boyce Principal Investigator, HMR

Place - Yves GiLLON
Head . Karen Dequatre Cheeseman
Trumple trend Clinical Project Manager
Sciences DNDi
DND

Robert Don Head of Filarial Diseases Program DNDi City 2 na 2017

Signature Date Date

Signature — 16 March 2017
Date

Signature

### 3 Introduction

This Statistical Analysis Plan (SAP) is based on the current trial protocol (version 5, Final 18 January 2017). Where statistical methods differ substantially between this SAP and the protocol, the differences will be identified in the SAP.

This SAP describes the datasets and the statistical methods to be used for the reporting and analysis of all data collected in Part 2 (cohorts 9 and 10), except for the 12-lead ECG continuous monitoring data which will be analysed by iCardiac Ltd (or an alternative provider), if applicable.

The randomisation code will not be broken before this SAP is finalised and signed. If a future protocol amendment necessitates a substantial change to the statistical analysis of the trial data, this SAP will be amended accordingly. If, after database lock, additional analyses are required to supplement the planned analyses described in this SAP, those unplanned analyses will not be described in an amended SAP, but they will be identified in the integrated clinical trial report (CTR). Any deviations from this SAP will be documented in the CTR.

This SAP has been written in consideration of the following guidelines:

- International Conference on Harmonization (ICH) E9, Guidance for Industry: Statistical Principles for Clinical Trials (ICH E9 1998)<sup>1</sup>; and
- ICH E3, Guidance for Industry: Structure and Content of Clinical Study Reports (ICH E3 1995)<sup>2</sup>.

Pharmacokinetic analysis will be done using WinNonlin v6.3 on a Windows PC. Statistical analysis will be done using SAS<sup>®</sup> 9.3 on a Windows PC.

# 4 Study Objective(s) and Endpoint(s)

### 4.1 Study Objective(s)

### 4.1.1 Primary Objective(s)

• To investigate the safety and tolerability of emodepside (BAY 44-4400) after single oral doses administered as solution or immediate release (IR) tablets in healthy male subjects.

### 4.1.2 Secondary Objective(s)

• To investigate the pharmacokinetics (PK) of emodepside (BAY 44-4400), after administration as oral solution, and IR tablet (optional)

- To conduct an exploratory investigation of the relative bioavailability of the 5 mg and 20 mg IR tablet formulation using data generated in this study (optional)
- Possibility to determine the effect of food on the bioavailability of emodepside (BAY 44-4400) after single oral doses administered as solution or IR tablets.

## 4.2 Study Endpoint(s)

### 4.2.1 Safety and Tolerability Variables:

- Adverse Events (AEs).
- Physical and Neurological examination findings (including assessments of alertness, speech, language, and comprehension; cranial nerves; motor exam; coordination/cerebellar function; tremor of the hands, legs and head (postural, kinetic and rest tremor); sensation; and gait and postural stability (Pull test); mood; and sleepiness.).
- Vital signs: heart rate (HR), systolic and diastolic blood pressure (BP) in supine and sitting position (Cohort 10 only in supine), weight, body mass index (BMI; height at screening only), oral temperature.
- 12-lead ECG (HR, PR, QRS, QTcF), and for selected cohorts 12-lead ECG continuous recording (for emodepside exposure response analysis HR, PR, QRS and QTcF).
- Clinical laboratory parameters:
   <u>Hematology</u>: hemoglobin, hematocrit, MCV, MCH, MCHC, platelets, reticulocytes, white blood cells (WBC) differential, red blood cells (RBC), glycated haemoglobin (HbA1C) (at screening);
  - <u>Coagulation</u>: activated partial thromboplastin time (aPTT), prothrombin time (PT);
- <u>Biochemistry</u>: aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP), glutamate dehydrogenase (GLDH), gamma-glutamyl transpeptidase (GGT), LDH, CK, amylase, lipase, free T4 and T3, thyroid-stimulating hormone (TSH), glucose, cholesterol (high-density lipoprotein [HDL], and low-density lipoprotein [LDL], total), triglycerides, creatinine, urea, uric acid, bilirubin (total and conjugated), total protein, sodium, potassium, calcium, chloride and magnesium in serum;

• <u>Urinalysis</u>: by dipstick - glucose, ketone bodies, specific gravity, occult blood, pH, proteins, leucocytes, bilirubin, urobilinogen, nitrites.

• Ophthalmological assessments (Cohort 10 only)

#### 4.2.2 Pharmacokinetic Variables:

Based on the plasma concentration time data, the following PK parameters of emodepside will be calculated.

- Main PK parameters: AUC<sub>∞</sub>, AUC<sub>∞</sub>/D, C<sub>max</sub>, C<sub>max</sub>/D, of emodepside (BAY 44-4400)
- Exploratory PK parameters:  $C_{max,norm}$ ,  $T_{max}$ ,  $t_{1/2}$ , MRT, CL/F,  $AUC_{\infty,norm}$ ,  $AUC_{t}$ ,  $AUC_{t,norm}$ ,  $V_{z}/F$  of emodepside (BAY 44-4400)
- Other parameters:  $\lambda_z$ ,  $AUC_{t-\infty}$ , points terminal

The following PK parameters of metabolites of emodepside may be calculated:  $AUC_{\infty}$ ,  $AUC_{\infty}/D$ ,  $C_{max}$ ,  $C_{max}/D$ ,  $C_{max,norm}$ ,  $T_{max}$ ,  $T_{1/2}$ ,  $AUC_{\infty,norm}$ ,  $AUC_{t}$ ,  $AUC_{t,norm}$ 

In urine, the amount and concentration of emodepside and possibly its metabolites will be measured. The appropriate specific PK parameters to be calculated will be decided according to the concentration.

### 4.2.3 Pharmacodynamic Variables:

- Profiles of glucose and insulin, glucagon and cortisol (Cohort 9 only), only on Pre-Day (Day -1), Profile Day (Day 0), and Day 1.
- Single samples of prolactin and leptin, only on Pre-Day (Day -1), Profile Day (Day 0), and Day 1(Cohort 9 only).

# 4.3 Statistical Hypotheses

No formal statistical testing will be done.

# 5 Study Design

This is a single-center, blinded, randomised, placebo-controlled, parallel-group, single-dose, 2-cohort, dose-escalation, comparison study investigating safety, tolerability, and PK of

emodepside, after administration as an oral liquid service formulation (LSF) solution in healthy male subjects. Within each cohort, subjects will be randomised to receive either emodepside or placebo (n=8 per cohort; 6 assigned to emodepside and 2 assigned to placebo).

Subjects in Cohort 9 will receive 10mg solution of emodepside or matching placebo in a fed state and subjects in Cohort 10 will receive 40mg solution of emodepside in fasted state.



**Table 1: Time and Events Table (Part 2, Cohort 9)** 

| Study Procedure | Screen | | | | | | | | | | | | | | | In-P | atien | t Pha | ise <sup>a</sup> | | | | | | | | | | | | | | | T | able <sup>b</sup> | Fo | llow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | | | | | | Pre | -Day | | | | | | | | | | Pro | file-l | Day | r | | | | | | | Eva | luat | ion | | | 3 | ee 12 | ible " | | Up |
| Day<br>± allowable deviation | -28 to -2 | -2 | | | | | • | 1 | | | | | | | | | | | 0 | | | | | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | | | | | 7<br>+3 |
| Subject information and Informed Consent | Х | | | | | | | | | | | | | | | | | | | | | | | | | 6 | | | | | | | | | | | |
| Medical history (including demographics and previous / concomitant medications) | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical examination <sup>c</sup> | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | Χ |
| Neurological examination <sup>d</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | Χ |
| Ward Admission (approx.16h) | | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Urine drugs of abuse and alcohol breath test | Х | Χ | | | | | | | | | | | | | | | | | | | | ) | | | | | | | | | | | | | | | |
| Hours <sup>a</sup> (pre/post drug) | | -36 | -24° | -23.5 | -23 | -22. | -22 | -21 | -20 | -18 | -16 | -12 | 0* | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 5 | 6 | 8 | 12 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | | | | | |
| Glucose, Insulin, Glucagon, and Cortisol profiles | | | Х | | Х | | Х | | Χ | | | X | Х | | X | • | Х | | | Х | | | | Χ | Χ | | | | | | | | | | | | |
| Samples for Prolactin & Leptin | | | Х | | | | | | | | | | Х | | | | | | | | | | | | Χ | | | | | | | | | | | | |
| Administration of emodepside <sup>e</sup> | | | | | | | | | | | | | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| 12-lead safety ECG <sup>f</sup> | Х | | X <sup>f</sup> | Χ | Χ | Х | Х | Χ | X | | Χ | X | Χ <sup>f</sup> | Χ | Χ | Χ | Χ | | Χ | Х | | | Χ | Χ | Х | | Χ | Χ | Χ | Χ | Χ | Χ | | | | | Χ |
| ECGs extracted from continuous recordings <sup>9</sup> | | | | | | | | | | | | | Xa | Xg | Xg | Xg | Χg | Χg | Xg | Χ <sup>g</sup> | | Χg | Xg | Χ <sup>g</sup> | Xg | | | | | | | | | | | | |
| Vital signs <sup>h</sup> | Х | | X <sup>h</sup> | Χ | Х | Х | Xh | Х | Xh | Х | X | X <sup>h</sup> | Xh | X | Χ | Χ | Χ <sup>h</sup> | | Χ | Xh | | Χ | Χ | Χ <sup>h</sup> | $\chi^h$ | | Χ | | | Χ | Χ | Х | | | | | Χ |
| Adverse event monitoring | Х | Χ | Χ | | | | Χ | | X | | | X | Х | | Χ | | Χ | | Χ | Χ | | Х | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | | | | | Χ |
| PK and metabolites <sup>j</sup> in plasma | | | | | | | | | | | | | X <sup>j</sup> | Х | X <sup>j</sup> | Χ | X <sup>j</sup> | Χ | Χ | X <sup>j</sup> | | Х | X <sup>j</sup> | X <sup>j</sup> | X <sup>j</sup> | Х | $X^{j}$ | Χ | Х | Х | Χ | Х | | | | | Х |
| PK in urine <sup>k</sup> | | | | | | | | | | | | | | | | 0-4 <sup>k</sup> | | | | | 4–8 <sup>k</sup> | • | 8-12 <sup>k</sup> | 12-24 <sup>k</sup> | | | | | | | | | | | | | |
| Laboratory Safety <sup>l,m</sup> | X m | | Χ | | | | | | | | | | Χ | | | | | | | | | | | | Χ | | Χ | Χ | Χ | Χ | Χ | Х | | | | | Χ |
| Neurological <sup>d</sup> examination and short physical examination <sup>c</sup> | | | Xc | | | | Х | | Х | | | Х | Х | | | | Х | | | Х | | | | Х | Х | Х | Х | | | | | | | | | | |

<sup>\*:</sup> In fasted subjects, all assessments at Hour –24 on Day –1 and Hour 0 on Day 0 are immediately before the administration of study drug (emodepside). In fed subjects, all assessments at Hour –24 on Day –1 and at Hour 0 on Day 0 are before the FDA breakfast. The only exception is the 12-lead ECG continuous recording (see footnote g).

<sup>&</sup>lt;sup>a</sup>: Including a 10-minute supine phase before supine BP, HR, body temperature, ECG; and for 5 minutes after each nominal timepoint for ECGs extracted from continuous recording (see footnote); and also recommended before drawing blood samples. Before sitting BP assessments minimum 3-minute sitting period.

b: If mean half-life of emodepside in any cohort is longer than predicted, there are options to extend in-house period, or out-patient ambulatory visits up to Day 14 if necessary, from Cohort 5 onwards and in subsequent cohorts. Refer to Option 1, Option 2, and Option 3 as outlined in Table .

Sponsor code: DNDI-EMO-001 Part 2

- c: Height at screening only, for calculation of BMI. Weight at screening for calculation of BMI, also at -24h (Day -1) for PK calculations.
- d: Neurological examination designed for the study, see Protocol Section 8.19.4 and Study Procedures Manual
- e: Administration of study drug while fasting or after a high-calorie, high-fat breakfast
- f: To include 3 repeat ECGs at these timepoints, with a time difference of about 1 minute, and single recordings at other timepoints
- <sup>9</sup>: For selected cohorts in Part 1 (see Protocol Section 8.19.2 continuous 12-lead ECG recording will be started 1 hour before dosing and continue for 24 hours post-dosing. ECGs will be extracted at predose, at three timepoints (-60, -45, and -30 minutes for fasted subjects or -90, -75, and -60 minutes for fed subjects) and at the timepoints at which PK blood samples are drawn. Subjects will be supine for 10 minutes prior to and 5 minutes after each nominal timepoint. When ECG extraction coincide with safety ECGs, vital signs and blood draws, procedures will be performed in said order.
- h: Vital signs to include BP (supine; plus sitting BP at the indicated timepoints<sup>th</sup>) and HR. Oral temperature only at screening and -24h.
- . Adverse Event (AE) monitoring will be throughout the study (spontaneous and solicited) to include questioning for tolerability and safety, however at these indicated timepoints will be specific questioning about AEs.
- In addition to the PK sample, metabolite samples are collected only for the indicated time points <sup>1</sup>. As an option, at the sponsor's discretion, an additional sample of no more than 1mL may be taken at each PK timepoint from all subjects in up to 2 cohorts.
- k: Start and end of urine collection for each bottle are indicated as hours post drug...
- Hematology, Coagulation, Chemistry: Urinalysis by dip stick.
- ": At Screening only: HIV 1, 2, Hepatitis B, C, HbA1C, in additional to hematology, coagulation, urinalysis, and chemistry.

Table 2. Follow-Up after Day 7 – Schedule Options 1, 2, or 3 Depending on Emodepside Plasma Concentrations at Day 7 in Previous Cohort(s) (from Cohort 5 onwards), Respectively.

For Screening and Days -2 through Day 8 see Table 1

| | T | | | | | |
|---|---|---|---|---|---|---|
| OPTION 1 | | | | Out-Patient Phase | | |
| Day | | | | | | Follow-Up Visit |
| | Discharge on Day 7 | | • | | | at 3 weeks (+3 days) post-dose |
| Physical Examination | , , | | | | | (see Table 1) |
| Neurological Examination | | | | | | (see Table 1) |
| 12-lead ECG | | | | | | (see Table 1) |
| Vital signs <sup>h</sup> | | | | | | (see Table 1) |
| Adverse event monitoring | | | | | | (see Table 1) |
| PK in plasma | | | | | | (see Table 1) |
| Laboratory Safety <sup>l,m</sup> | | | | | | (see Table 1) |
| OPTION 2 | | | | <b>Out-Patient Phase</b> | | |
| Day | Un to A via | to duni | ing the national from Day 9, 21 in | alusiya (as noodad) | | Follow-Up Visit |
| Day | - | | ing the period from Day 8–21 inc | clusive (as needed) | | at 3 weeks (+3 days) post-dose |
| N : 15 | Ambulatory Evaluation Visits, S | chedul | led As Needed | | | |
| Physical Examination | | | | | | (see Table 1) |
| Neurological Examination | | | | | | (see Table 1) |
| 12-lead ECG | | | | | | (see Table 1) |
| Vital signs <sup>h</sup> | | | | | | (see Table 1) |
| Adverse event monitoring | X | | X | X | X | (see Table 1) |
| PK in plasma | X | | X | X | X | (see Table 1) |
| Laboratory Safety <sup>l,m</sup> | X | | X | X | X | (see Table 1) |
| OPTION 3 | | | Discharge from Ward on Day | ΥX | | |
| _ | 8 (±1) | | 10 (±1) | 12 (±2) | 14 (±2) | |
| Day | (as needed) | | (as needed) | (as needed) | (max.) | Follow-Up Visit |
| | Prolonged In-House Evaluation | Phase | | / | | at 3 weeks (+3 days) post-dose |
| | with Discharge from Ward on D | | | | | are means (ve auje, peer acce |
| Physical Examination | | | | | | (see Table 1) |
| Neurological Examination | | | | | | (see Table 1) |
| 12-lead ECG | | | | | | (see Table 1) |
| Vital signs <sup>h</sup> | | | | | | (see Table 1) |
| Adverse event monitoring <sup>i</sup> | X | | X | Χ | X | (see Table 1) |
| PK in plasma | X | | X | X | X | (see Table 1) |
| Laboratory Safety <sup>l,m</sup> | X | | X | X | X | (see Table 1) |

Table 3. Schedule of Events (Part 2, Cohort 10)

| Study Procedure | | ening<br>sits | | | | | | | | | | | | In-Patient Phase <sup>a</sup> | | | | | | | | | | | | | | | t-pati | | Follo | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 1 | 2 | | | | | | Pre | -Da | у | | | | | | | | | Pro | ofile- | Day | | | | | | | I | Eva | luat | ion | | | ı | ohase | ' | w-Up |
| Day ± allowable deviation | -28 to<br>-2 | -7 to<br>-1 | -2 | | | | | | -1 | | | | | | | | | | | 0 | | | | | | | | 2 | 3 | 4 | 5 | 6 | 7 | 10<br>±1 | 14<br>±2 | 18<br>±2 | 21<br>+3 |
| Subject information and Informed Consent | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Medical history<br>(including<br>demographics,<br>previous/concomitant<br>medications) | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical examination <sup>b</sup> | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | Χ |
| Neurological examination <sup>c</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | Х |
| Colour blindness test <sup>d</sup> | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Ophthalmology exam <sup>e</sup> | | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | ı |
| Ward Admission (approx.16h) | | | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Urine drugs of abuse and alcohol breath test | Х | | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Hours <sup>a</sup> (pre/post<br>drug) | | | -36 | -24* | -23.5 | -23 | -22.5 | -22 | -21 | -20 | -18 | -16 | -12 | 0* | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 5 | 6 | 8 | 12 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | | | | |
| Glucose and Insulin profiles | | | | Х | | Х | | | | | | | X | X | | Х | | | | | | | | | Χ | Х | | | | | | | | | | | |
| Administration of emodepside <sup>f</sup> | | | | | | | | | | | | * | | Х | | | | | | | | | | | | | | | | | | | | | | | |
| 12-lead safety ECG | Х | | | Χg | | Χ | | | | | | | X | Χ <sup>g</sup> | | Χ | | | | | | | | | Χ | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | | | | Χ |
| Vital signs <sup>h</sup> | Χ | | | Χ | Χ | Χ | | | | | | X | Χ | Х | Χ | Χ | | | | | | | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | | | Χ |
| Adverse event monitoring <sup>i</sup> | Х | | Х | Х | | | | X | | X | | | X | Х | | Х | | Χ | | Х | Χ | | Χ | Х | Х | Х | Х | Χ | Х | Χ | Х | Χ | Х | Х | Х | Χ | Х |
| PK in plasma <sup>j</sup> | | | | | | | | | | | | | | Х | Χ | Χ | | | | (X) | | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ |
| Laboratory Safety <sup>k,l</sup> | Χ <sup>I</sup> | | | Χ | | | | | 1 | | | | | Х | | | | | | | | | | | | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Х |
| Neurological <sup>c</sup> examination and short physical examination <sup>b</sup> | | | | X <sub>p</sub> | | Х | | | | | | | Х | Х | | Х | | | | | | | | | Х | Х | х | Х | | | | | | | | | |
| Travel and stay at ophthalmology clinic | | | | | | | | | | | | | | | | | Χ | Χ | Χ | Х | Χ | Х | | | | | | | | | | | | | | | |
| Ophthalmology exam <sup>m</sup> | | | | | | | | | | | | | | | | | | | Χ | | | | | | | | | | | | | | | | <u> </u> | | |

<sup>\*</sup> All assessments at Hour 0 on Day 0 are immediately before the administration of study drug (emodepside), and assessments at Hour –24 on Day –1 will be time-matched to Profile Day

HMR code: 15-020 Part 2

Sponsor code: DNDI-EMO-001 Part 2

(dosing Day)

a Including a 10-minute supine phase before supine BP, HR, body temperature, ECG; and also recommended before drawing blood samples.

b Height at screening only, for calculation of BMI. Weight at screening for calculation of BMI, also at -24h (Day -1) for PK calculations.

<sup>&</sup>lt;sup>c</sup> Neurological examination designed for the study, see Protocol Section 8.19.4 and Study Procedures Manual.

<sup>&</sup>lt;sup>d</sup> Colour blindness to be determined at Screening visit 1.

e If subjects are eligible for study entry based on Screening visit 1 assessments, they will be asked to undergo an ophthalmology exam (Screening visit 2) within a week before Profile Day or on Pre–Day at the latest. All assessments for Screening Visit 1 will be performed prior to Screening Visit 2, but visits can be combined if necessary.

f Administration of study drug is in the fasted-state only.

<sup>&</sup>lt;sup>9</sup> To include 3 repeat ECGs at these timepoints, with a time difference of about 1 minute, and single recordings at other timepoints.

<sup>&</sup>lt;sup>h</sup> Vital signs to include supine BP and HR. Oral temperature only at screening and -24h.

Adverse Event (AE) monitoring will be throughout the study (spontaneous and solicited) to include questioning for tolerability and safety, however at these indicated timepoints will be specific questioning about AEs.

<sup>&</sup>lt;sup>j</sup> Timepoint shown as (X) indicates sample will be taken off-site whilst at the ophthalmology clinic. As an option, at the sponsor's discretion, an additional sample of no more than 1 mL may be taken at each PK timepoint from all subjects in up to 3 cohorts.

<sup>&</sup>lt;sup>k</sup> Hematology, Coagulation, Chemistry; Urinalysis by dip stick.

At Screening only: HIV 1, 2, Hepatitis B, C, HbA1C, in additional to hematology, coagulation, urinalysis, and chemistry.

<sup>&</sup>lt;sup>m</sup> Ophthalmology exams will be performed on Profile-Day (Day 0) approximately 2-2.5 h post-dose. If deemed necessary by the ophthalmologist additional ophthalmology follow-up visit(s) may be scheduled for eve-related AEs.

# 6 Planned Analyses

### 6.1 Interim Analyses

No interim analyses are planned. However, the blinded safety and PK data will be reviewed after Cohort 9.

#### **6.1.1** Persons responsible for analysis

Toni Mitchell (HMR) Statistician

Nick Jackson (HMR) SAS Programmer

## 6.2 Final Analysis

The database will be locked once all subjects have completed the study, data have been entered and all queries resolved. The final analysis will be carried out following database lock and unblinding.

#### 6.2.1 Persons responsible for analysis

Stephen Sah (HMR) Statistician

Nick Jackson (HMR) SAS Programmer

Bhavini Ladwa (HMR) Data Manager

# 7 Sample Size Considerations

# 7.1 Sample Size Assumptions

No formal sample size calculations have been performed as this is an exploratory study. A sample size of 8 per cohort will be considered sufficient to examine the safety and tolerability of emodepside as well as the PK after single oral administration of the investigational drug. For evaluation, a minimum number of 6 evaluable subjects per cohort is required.

HMR code: 15-020 Part 2

Sponsor code: DNDI-EMO-001 Part 2

# 8 Analysis Populations

The following population sets will be identified:

Safety Population: All subjects who received at least one dose of IMP.

PK Concentration Population: All subjects who received at least one dose of IMP and for

whom a pharmacokinetic sample has been analysed.

PK Parameter Population: All subjects in the PK Concentration Population for whom

pharmacokinetic parameters can be derived.

In all populations, treatment will be assigned based upon the treatment subjects actually received, regardless of the treatment to which they were randomised.

The primary endpoint will be analysed using the safety population.

## 8.1 Analysis Datasets

All analysis datasets will be based on observed data, except as outlined in Section 10.2.

## 9 Treatment Comparisons

The treatment comparison of interest is active (emodepside) versus placebo.

## 9.1 Data Display Treatment and Other Subgroup Descriptors

The sort order for treatment groups will be placebo, then study treatment in ascending dose order.

Listings of data will be sorted and displayed by treatment group, subject number, and also by date and time if applicable.

All subjects in cohorts 9 and 10 receiving the same formulation of placebo will be combined to form a pooled placebo group.

The treatment descriptions to be used on all tables and listings are:

Treatment GroupsShort DescriptionPlacebo [solution](Fed)PLA [sol](Fed)Placebo [solution](Fasted)PLA [sol](Fasted)Emodepside (xx mg) [solution](Fed)xx mg [sol](Fed)Emodepside (xx mg) [solution](Fasted)xx mg [sol](Fasting)

#### 9.1.1 Conventions for Summary Statistics and Data Displays

The minimum set of summary statistics for numeric variables will be: n, mean, standard deviation (or standard error), median, minimum, and maximum. 95% confidence intervals will be presented where appropriate for data interpretation.

Categorical data will be summarised in frequency tables with n and percentage. Summaries of a categorical variable will include all recorded values.

The minimum and maximum values will be presented with the same number of decimal places as the raw data collected on the CRF (or to 3 significant figures for derived parameters). The mean and percentiles (e.g. median, Q1, and Q3) will be presented using one additional decimal place. The standard deviation and standard error will be presented using two additional decimal places.

Placebo subjects will be pooled across cohorts 9 and 10 taking into account formulation and fed/fasted status.

## 10 Data Handling Conventions

### 10.1 Premature Withdrawal and Missing Data

All subjects who withdraw prematurely from the study or study drug will be included in the statistical analyses.

If a subject completes the treatment period but has missing data, then this will be made apparent in the subject listings. Missing data will not be imputed except for as outlined in Section 10.2.

If the study is prematurely discontinued, all available data will be listed and a review will be carried out to assess which statistical analyses are still considered appropriate.

Data collected at unscheduled time points during the study will not be used in the summaries or data analyses. They will be included in the listings.

If time information (i.e. hours and/or minutes) for adverse events or concomitant medication is missing, but the day is present, then the time will be calculated in days. If date information is partial or missing, then any derived times (e.g. AE start time from last study medication) will be listed as missing.

Conventions for handling missing plasma concentrations are given in Appendix B.

#### 10.2 Derived and Transformed Data

For ECGs, vital signs, glucose, insulin, glucagon, cortisol and neurological examinations recorded on Day -1 the baseline will be the -24 h value and for Day 0 the baseline will be the pre-dose value on Day 0. The AUC<sub>0-24</sub> for change from baseline in glucose, insulin, glucagon and cortisol will be calculated on Day -1 and Day 0, using the linear-linear trapezoidal method. For prolactin and leptin the baseline will be pre-dose on Day 0.

Laboratory data will be reported in standard units. The baseline will be the latest value recorded pre-dosing on Day 0. Out-of-range laboratory tests may be repeated. If a test is out-of-range at a baseline timepoint and repeated before dosing, the latest repeat value before dosing will be used as baseline. However, if a test is out-of-range and repeated at any other time during the study, the out-of-range value (not the repeat value) will be included in statistical summaries.

Triplicate ECG measurements will be made at some timepoints on Day -1 and Day 0, the mean of the three measurements for each subject will be used at each timepoint.

The pharmacokinetic parameters to be derived are given in Appendix B

#### 10.3 Assessment Windows

No assessment windows are defined for this report.

### 10.4 Values of Potential Clinical Importance

Any laboratory value outside the reference interval for that variable will be flagged with an 'H' if it is higher than the reference interval, and with an 'L' if it is lower. Additionally, if, during the course of the trial, a variable changes from baseline (Day 0) by more than a predetermined amount (as defined by the Principal Investigator, Appendix A), that value will receive a flag 'I' if increased, or 'D' if decreased. Therefore, if a value both falls outside the reference interval and alters from the baseline value by more than the predetermined amount, it will attract a double flag and will be considered to be potentially clinically important.

A vital signs result will be considered to be of potential clinical importance if it falls outside the relevant range below:

| Vital Sign | Range |
|------------------------------------------------|------------------|
| Supine/semi-recumbent systolic blood pressure | 85–160 mm Hg |
| Supine/semi-recumbent diastolic blood pressure | 40–90 mm Hg |
| Supine/semi-recumbent heart rate | 40–100 beats/min |
| Respiration rate | 8–20 per min |
| Oral temperature | 35.5–37.8°C |

QTcB or QTcF > 450 msec and increases in QTcB or QTcF from baseline of > 30 msec will be considered to be potentially clinically important.

# 11 Study Population

## 11.1 Disposition of Subjects

The disposition of all subjects in the safety population will be summarised including: number of subjects randomised; number completing the study (i.e. not withdrawn), by treatment; and number discontinued (withdrawn) from the study. The number of subjects in each analysis population will be summarised by treatment.

All subjects who withdraw or are withdrawn from the study will be listed, by treatment, with the reason for withdrawal.

A listing of analysis populations will be provided.

#### 11.2 Protocol Deviations

Before closing the database, data listings will be reviewed to identify any significant deviations and determine whether the data should be excluded from any analysis populations.

Major protocol deviations include subjects who:

- Entered the study even though they did not satisfy the entry criteria.
- Met the criteria for withdrawal from the study but were not withdrawn.
- Received the wrong treatment or incorrect dose.
- Received an excluded concomitant therapy.
- Received investigational product(s) past the expiration date and time.

• Had their treatment assignment unblinded.

In addition, subjects with minor time deviations (measurements taken outside the allowable windows given in the protocol) will be identified.

### 11.3 Demographic and Baseline Characteristics

Demographic and baseline characteristics (e.g. physical examination, neurological examination, vital signs and ECGs) will be listed and summarised.

Subjects who take concomitant medication will be listed. All non-trial medication will be coded using version September 2016 of the WHO Drug dictionary.

### 11.4 Treatment Compliance

Dates and times of dosing will be listed.

# 12 Safety Analyses

Summaries and listings of safety data will use the safety population.

## 12.1 Extent of Exposure

The dates and times of treatment dosing will be listed to indicate exposure to the study medication.

#### 12.2 Adverse Events

Adverse events will be coded using the version of the Medical Dictionary for Regulatory Activities (MedDRA) (version 20.0).

All adverse events will be listed.

The number of subjects with at least one treatment-emergent adverse event (TEAE) will be tabulated by actual treatment and MedDRA system organ class and preferred term. A treatment-emergent adverse event is defined as an event emerging during treatment having been absent pre-treatment or having worsened relative to pre-treatment.

For each of the following, the number of subjects with adverse events will be summarised by actual treatment:

• TEAEs by system organ class and preferred term

• Drug-related ("related" as recorded by the Investigator) TEAEs by system organ class and preferred term

Subjects with more than one TEAE will be counted only once, at the greatest severity or causal relationship, for each system organ class and preferred term. Adverse events with missing severity and/or causality will be treated as severe and related, respectively.

Summaries will be sorted by system organ class and decreasing total incidence of preferred term.

#### 12.3 Deaths and Serious Adverse Events

Adverse events leading to deaths and serious adverse events will be listed separately (fatal events will be listed separately from non-fatal events).

### 12.4 Adverse Events Leading to Withdrawal from the Study

Adverse events leading to withdrawal will be listed separately.

### 12.5 Clinical Laboratory Evaluations

Haematology, clinical chemistry and urinalysis evaluation at each planned assessment, and change from baseline at each planned post-baseline assessment, will be summarised by actual treatment.

Urinalysis parameters will also be listed.

All laboratory values of potential clinical importance will be listed and all related laboratory results (i.e. haematology or clinical chemistry) for subjects with values of potential clinical importance will be listed, separately. Frequencies of laboratory values of potential clinical importance will be summarised.

## 12.6 Other Safety Measures

#### 12.6.1 Vital signs

Vital signs evaluation at each planned assessment, and change in vital signs baseline at each planned post-baseline assessment, will be summarised by actual treatment. Individual subject profiles will be plotted for each vital sign parameter (Blood Pressure and Heart Rate).

Vital signs data of potential clinical importance will be listed separately.

#### 12.6.2 ECG

QT interval data will be presented using Bazett's (QTcB) and Fridericia's (QTcF) corrections.

ECG data will be summarised by treatment and time point. Differences from baseline will be summarised by treatment and time point.

The number of subjects with a potentially clinically important ECG value will be summarised by actual treatment and time point, giving the numbers of subjects with QT, QTcB or QTcF > 450 msec, > 480 msec and > 500 msec, and the numbers of subjects with increases in QT, QTcB or QTcF from baseline of > 30 msec and > 60 msec<sup>3</sup>. A supporting listing of all subjects with an ECG value of potential clinical importance and a separate listing of ECG findings classified as abnormal by the Investigator will also be provided.

### 12.6.3 Neurological examination

Neurological examination results will be summarised and normal and abnormal neurological examination findings will be listed in detail according to the CRF. Total scores from neurological questionnaires at each planned assessment, and change from baseline at each planned post-baseline assessment, will be summarised by actual treatment.

Total scores from neurological questionnaires will also be listed.

## 12.6.4 Physical examination

Physical examination results will be summarised and abnormal physical examination findings will be listed.

#### 12.6.5 Ophthalmology assessments

Ophthalmology assessments results will be summarised and listed by time point.

# 13 Pharmacokinetic Analyses

Analytical Services International Ltd, London, U.K. will measure the plasma and urine concentrations of emodepside. The pharmacokinetic analysis will be done by Statistics and Data Management Department at HMR. Pharmacokinetic parameters will be calculated using WinNonlin, version 6.3.

In addition, the plasma and urine concentration of emodepside metabolite(s) may be measured. If and when these data become available a SAP amendment will be written to specify their reporting (if applicable).

The pharmacokinetic parameters to be derived are given in Appendix B.

PK concentration data will be summarised using the PK concentration population. PK parameters will be summarised using the PK Parameter population.

For log transformed parameters, the primary measure of central tendency will be the geometric mean<sup>4</sup>; for untransformed parameters, it will be the arithmetic mean or median.

For all variables N (number of subjects receiving the treatment/formulation in the population), n (number of observations), arithmetic mean, median, minimum, maximum, SD, %CV, and the 95% confidence interval for the arithmetic mean will be provided. For log-transformed variables, all of the above plus the geometric mean, which is the anti-logged arithmetic mean of log-transformed variables, its 95% confidence interval and the SD of the logs will be provided.

The between-subject CV will be calculated using:

- 1. %CVb = 100 \* (SD/Mean) with SD and Mean of untransformed data
- 2. %CVb =  $100 * \sqrt{(\exp(SD)^2 1)}$  with SD of log-transformed data

### 13.1 Plasma PK

#### 13.1.1 Pharmacokinetic Concentration Data

The plasma concentrations of emodepside and metabolites (if applicable) will be listed and summarised by treatment. Means at any time will only be calculated if at least 2/3rds of the individual data points are above the lower limit of quantification.

Individual and mean plasma concentration—time profiles will be presented graphically.

#### 13.1.2 Pharmacokinetic Parameters

The pharmacokinetic parameters of emodepside and metabolites (if applicable) will be listed and summarised by treatment.

To assess the effect of food, analysis of variance (ANOVA) models will be fitted to the fed (Part 2, Cohort 9) solution and relevant fasted (Part 1, Cohort 5) solution data with the logarithm of the pharmacokinetic parameters  $AUC_{0-24}$  as the dependent variable, and formulation as a fixed effect. The estimated least square means and residual variance from the model will be used to construct 90% CIs for the difference in means on the log scale for the comparison of fed versus fasted solutions.

## 13.2 Urinary PK

If concentrations of emodespide in urine are determined, the amount of emodespide excreted in the urine will be estimated. The data will be listed and summarised by treatment.

# 14 Pharmacodynamic Analyses

Summaries and listings will use the safety population.

Pharmacodynamic variables (glucose, insulin, glucagon, cortisol, prolactin and leptin) at each planned assessment, and change from baseline at each planned post-baseline assessment, will be summarised by actual treatment.

In addition, for glucose and insulin (Cohorts 9 and 10), glucagon and cortisol (Cohort 9):

- Individual subject profiles will be plotted
- The difference between change from baseline on Day 0 and Day -1 will be summarised at each planned post-baseline assessment by actual treatment
- The AUC<sub>0-24</sub> of change from baseline will be summarised for each day and treatment

Individual Insulin and PK Concentration Plots, including Related Significantly Important AE Durations will be produced.

For calculation of pharmacodynamics parameters, summary statistics and individual profile plots, values below the quantifiable limit of the assay will be substituted by one half of the lower limit of quantification.

# 15 Changes from the Protocol Specified Statistical Analysis

After the study was submitted to the MHRA and ethics committee the following changes were made to the analyses:

- 1) The definition of treatment-emergent adverse event has been updated from "an AE will be considered as treatment emergent if it appeared after the first dosing, or if appeared before dosing and worsened after dosing" to:
  - A treatment-emergent adverse event is defined as an event emerging during treatment having been absent pre-treatment or having worsened relative to pre-treatment<sup>1</sup>.
- 2) The AUC<sub>0-24</sub> of change from baseline for glucose, insulin, glucagon and cortisol will be summarised for each day and treatment
- 3) The following emodepside parameters have been added to those mentioned in the protocol:

Main PK parameters: AUC<sub>0-24</sub> and AUC<sub>0-24</sub>/D

Exploratory PK parameters: AUC<sub>0-24</sub>,<sub>norm</sub> ,t<sub>1/2,dom</sub>

4) The following analyses have been added for glucose, insulin, glucagon and cortisol:

The difference between change from baseline on Day 0 and Day -1 will be summarised at each planned post-baseline assessment by actual treatment

The AUC<sub>0-24</sub> of change from baseline will be summarised for each day and treatment

#### 16 References

 International Conference on Harmonization, 1998. Statistical Principles for Clinical Trials - ICH Harmonised Tripartite Guideline. Guidance for Industry, E9, FDA federal register, Vol 63, 1998, p49583. Available at: http://www.fda.gov/cder/guidance.

2. International Conference on Harmonization, 1995. Structure and Content of Clinical Study Reports - ICH Harmonised Tripartite Guideline. Guidance for Industry, E3, FDA federal register, Vol 61, 1996, p37320. Available at: http://www.fda.gov/cder/guidance.

- International Conference on Harmonisation, 2005. Clinical Evaluation of QT/QTc
   Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs.
   Concept paper, Guidance for Industry, E14, Center for Drug Evaluation and Research (CDER). Available at: http://www.fda.gov/cder/guidance/6922fnl.htm.
- 4. Julious, SA & Debarnot, CAM (2000) "Why are Pharmacokinetic Data Summarised by Arithmetic Means?", Journal of Biopharmaceutical Statistics, 10 (1), p55-71.
- 5. FL140 HMR Laboratory alert and delta ranges ver 3 (HMR Lab form).

# 17 ATTACHMENTS

# 17.1 Table of Contents for Data Display Specifications

For overall page layout refer to Appendix C.

Tables, figures and listings will be labelled B for Part 2, e.g., 14.1B

The numbering in the tables below will take precedence over the numbering in the shells.



The following tables and figures will be produced (templates provided in Sections 17.2.1 and 17.2.2):

| Table | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 10.1 | Summary of Subject Disposition | Safety | 16.2.1.2,<br>16.2.3.1 | T_SD1 |
| 14.1 | DEMOGRAPHIC DATA | | | |
| 14.1 | Summary of Demographic Characteristics | Safety | 16.2.4.1 | T_DM1 |
| 14.2 | PHARMACOKINETIC AND PHARMACODYNAMIC DATA | | | |
| 14.2.1.1 | Summary of Emodepside Plasma Pharmacokinetic Concentration-Time Data (ng/mL) | PK | 16.2.6.1.1 | <u>T_PK1</u> |
| 14.2.1.2 | Summary of Derived Emodepside Plasma Pharmacokinetic Parameters | PK | 16.2.6.1.2 | <u>T_PK3</u> |
| 14.2.1.3 | Summary of Log-Transformed Derived Emodepside Plasma<br>Pharmacokinetic Parameters | PK | 16.2.6.1.2 | <u>T_PK4</u> |
| 14.2.1.4 | Assessment of the Effect of Food on the PK of Emodepside | PK | 16.2.6.1.2 | <u>T_PK7</u> |
| 14.2.2 | Summary of Derived Emodepside Urine Pharmacokinetic Parameters | PK | 16.2.6.2 | <u>T_PK3</u> |
| 14.2.3.1 | Summary of Glucose | Safety | 16.2.6.3 | <u>T_PD1</u> |
| 14.2.3.2 | Summary of Difference Between Day -1 and Day 0 in Glucose | Safety | 16.2.6.3 | <u>T_PD2</u> |
| 14.2.3.3 | Summary of AUC <sub>0-24</sub> for Change from Baseline in Glucose | Safety | 16.2.6.4 | <u>T_PD3</u> |
| 14.2.4.1 | Summary of Insulin | Safety | 16.2.6.3 | <u>T_PD1</u> |
| 14.2.4.2 | Summary of Difference Between Day -1 and Day 0 in Insulin | Safety | 16.2.6.3 | T_PD2 |
| 14.2.4.3 | Summary of AUC <sub>0-24</sub> for Change from Baseline in Insulin | Safety | 16.2.6.3 | <u>T_PD3</u> |
| 14.2.5.1 | Summary of Glucagon | Safety | 16.2.6.3 | <u>T_PD1</u> |
| 14.2.5.2 | Summary of Difference Between Day -1 and Day 0 in Glucagon | Safety | 16.2.6.3 | <u>T_PD2</u> |
| 14.2.5.3 | Summary of AUC <sub>0-24</sub> for Change from Baseline in Glucagon | Safety | 16.2.6.3 | T_PD3 |

| Table | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 14.2.6.1 | Summary of Cortisol | Safety | 16.2.6.3 | T_PD1 |
| 14.2.6.2 | Summary of Difference Between Day -1 and Day 0 in | Safety | 16.2.6.3 | <u>T_PD2</u> |
| | Cortisol | | | |
| 14.2.6.3 | Summary of AUC <sub>0-24</sub> for Change from Baseline in Cortisol | Safety | 16.2.6.3 | <u>T_PD3</u> |
| 14.2.7 | Summary of Prolactin | Safety | 16.2.6.3 | <u>T_PD1</u> |
| 14.2.8 | Summary of Leptin | Safety | 16.2.6.3 | <u>T_PD1</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Summary of Treatment-Emergent Adverse Events | Safety | 16.2.7.1 | T AE1 |
| 14.3.1.2 | Summary of Drug-Related Treatment-Emergent Adverse | Safety | 16.2.7.1 | T AE1 |
| | Events | | | |
| 14.3.1.3 | Summary of Treatment-Emergent Adverse Events by Severity | Safety | 16.2.7.1 | <u>T_AE1</u> |
| | Grade | | | |
| 14.3.1.4 | Summary of Drug Related Treatment-Emergent Adverse | Safety | 16.2.7.1 | <u>T_AE1</u> |
| | Events by Severity Grade | | | |
| 14.3.2.1 | Listing of Fatal Adverse Events | Safety | 16.2.7.1 | <u>L_AE1_PG</u> |
| 14.3.2.2 | Listing of Non-Fatal Serious Adverse Events | Safety | 16.2.7.1 | L_AE1_PG |
| 14.3.2.3 | Listing of Other Significant Adverse Events | Safety | 16.2.7.1 | L_AE1_PG |
| 14.3.3 | Narratives of deaths, other serious and significant adverse events | Safety | | - |
| 14.3.4 | Summary of Laboratory Values of Potential Clinical | Safety | 16.2.8.1, | <u>T_LB1</u> |
| | Importance | | 16.2.8.3 | |
| 14.3.5.1 | Summary of Chemistry Laboratory Values | Safety | 16.4 | <u>T_LB2</u> |
| 14.3.5.2 | Summary of Haematology Laboratory Values | Safety | 16.4 | T_LB2 |
| 14.3.5.3 | Summary of Urinalysis Dipstick Results | Safety | 16.2.8.5 | T_UR1 |
| 14.3.6.1 | Summary of Vital Signs | Safety | 16.4 | <u>T_VS1</u> |
| 14.3.6.2 | Summary of AUC0-24 for Change from Baseline in Supine Diastolic Blood Pressure (h*mmHg) | Safety | 16.4 | <u>T_VS2</u> |
| 14.3.6.3 | Summary of AUC0-24 for Change from Baseline in Supine Systolic Blood Pressure (h*mmHg) | Safety | 16.4 | <u>T_VS2</u> |
| 14.3.6.4 | Summary of AUC0-24 for Change from Baseline in Supine | Safety | 16.4 | T_VS2 |

| Table | Description | Population | Source<br>Listing | Template<br>(Shells below) |
|---|---|---|---|---|
| | Heart Rate (h*beats/min) | | | |
| 14.3.7.1 | Summary of ECG values | Safety | 16.4 | <u>T_EG2</u> |
| 14.3.7.2 | Summary of ECG Values and Changes in ECG Values of | Safety | 16.4 | T_EG3 |
| | Potential Clinical Importance | | | |
| 14.3.8.1 | Summary of Neurological Examination Data | Safety | 16.2.9.5 | T_NE1 |
| 14.3.8.2 | Summary of Neurological Examination Questionnaire Data | Safety | 16.2.9.6 | T LB2 |
| 14.3.9 | Summary of Physical Examination Data | Safety | 16.2.9.4 | T PE1 |
| 14.3.10 | Summary of Ophthalmological Examination Data | Safety | 16.2.9.7 | T NE1 |

| Figure | Description | Population | <b>Source Listing</b> | Template (Shells below) |
|---|---|---|---|---|
| 14.2 | PHARMACOKINETIC AND PHARMACODYNAMIC DATA | | | |
| 14.2.1.1 | Individual Emodepside Plasma Concentration-Time Plots (Linear and Semi-log) | PK | 16.2.6.1.1 | <u>F_PK1</u> |
| 14.2.1.2 | Geometric mean (+/- SD) Emodepside Plasma<br>Concentration-Time Plots (Linear and Semi-log) | PK | 16.2.6.1.1 | F_PK2 |
| 14.2.2.1<br>14.2.2.2 | Individual Glucose-Time Plots Individual Glucose and PK Concentration Plots - | PD<br>PD | 16.2.6.3<br>16.2.6.3, | <u>F_PD1</u> |
| 11.2.2.2 | Including Related Significantly Important AE Durations | | 16.2.6.1.1,<br>16.2.7.1 | F_PD2 |
| 14.2.3.1 | Individual Insulin-Time Plots | PD | 16.2.6.3 | <u>F PD1</u> |
| 14.2.3.2 | Individual Insulin-Time Plots 0-12h | PD | 16.2.6.3 | <u>F_PD1</u> |
| 14.2.3.3 | Individual Insulin and PK Concentration Plots - | PD | 16.2.6.3, | F PD2 |
| | Including Related Significantly Important AE Durations | | 16.2.6.1.1, | |
| | | | 16.2.7.1 | |
| 14.2.4 | Individual Glucagon-Time Plots | PD | 16.2.6.3 | <u>F PD1</u> |
| 14.2.5 | Individual Cortisol-Time Plots | PD | 16.2.6.3 | <u>F PD1</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Individual Systolic Blood Pressure-Time Plots | Safety | 16.2.9.1 | F_PD1 |
| 14.3.1.2 | Individual Diastolic Blood Pressure-Time Plots | Safety | 16.2.9.1 | <u>F_PD1</u> |
| 14.3.2 | Individual Heart Rate-Time Plots | Safety | 16.2.9.1 | F_PD1 |

The following abbreviated listings will be produced (templates provided in Section 17.2.3):

| Listing | Description | Template (Shells below) |
|---|---|---|
| 16.2.1 | Study dates & disposition of subjects | , and the second |
| 16.2.1.1 | Listing of Study Dates | L SD1 PG |
| 16.2.1.2 | Listing of Reasons for Withdrawal | L SD2 PG |
| 16.2.2 | Protocol deviations | |
| 16.2.2.1 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | L DV1 PG |
| 16.2.2.2 | Listing of Subjects with Time Deviations | L_TD1_PG |
| 16.2.2.3 | Listing of Subjects with Other Protocol Deviations | L DV2 PG |
| 16.2.3 | Analysis sets, including subjects excluded from analysis | |
| 16.2.3.1 | Listing of Analysis Populations | L_AN1_PG |
| 16.2.4 | Demographic data & concomitant medication | |
| 16.2.4.1 | Listing of Demographic Characteristics | L DM1 PG |
| 16.2.4.2 | Listing of Concomitant Medications | <u>L_CM1_PG</u> |
| 16.2.5 | Study drug administration | |
| 16.2.5.1 | Listing of Exposure Data | <u>L_EX1_PG</u> |
| 16.2.6 | Pharmacokinetic and Pharmacodynamic data | |
| 16.2.6.1.1 | Listing of Emodepside Plasma Pharmacokinetic Concentration-Time | L PK1 PG |
| | Data | <u>LIKIIO</u> |
| 16.2.6.1.2 | Listing of Derived Emodepside Plasma Pharmacokinetic Parameters | <u>L_PK4_PG</u> |
| 16.2.6.1.3 | Individual Emodepside Plasma Concentration-Time Plots (log scale) for | F PK10 |
| | Estimation of λz, with Regression Line | <del></del> |
| 16.2.6.2 | Listing of Emodepside Urine Excretion Rate Data | L PK3 PG |
| 16.2.6.3 | Listing of PD concentration-Time Data | L PK1 PG |
| 16.2.6.4 | Listing of Derived AUC0-24 PD Concentration-Time Data | <u>L_PK1_PG</u> |
| 16.2.7 | Adverse events | |
| 16.2.7.1 | Listing of All Adverse Events | L_AE1_PG |
| 16.2.7.2 | Listing of Serious Adverse Events | L AE1 PG |

| 16.2.7.3 | Listing of Adverse Events Leading to Withdrawal from Study | L_AE1_PG |
|---|---|---|
| 16.2.8 | Laboratory values | |
| 16.2.8.1 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance | L_LB1_PG |
| 16.2.8.2 | Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities | L_LB2_PG |
| 16.2.8.3 | Listing of Haematology Abnormalities of Potential Clinical Importance | L LB1 PG |
| 16.2.8.4 | Listing of All Haematology Laboratory Data for Subjects with PCI Abnormalities | L_LB2_PG |
| 16.2.8.5 | Listing of Urinalysis Data | <u>L URI</u> |
| 16.2.9 | Vital signs, ECG variables, neurological, physical findings and Ophthalmological Assessment | |
| 16.2.9.1 | Listing of Vital Signs of Potential Clinical Importance | L VS1 PG |
| 16.2.9.2 | Listing of ECG Values of Potential Clinical Importance | L EG1 PG |
| 16.2.9.3 | Listing of Abnormal ECG Findings | L EG2 PG |
| 16.2.9.4 | Listing of Abnormal Physical Examination Findings | L PE1 PG |
| 16.2.9.5 | Listing of Neurological Examination Findings | L NE1 PG |
| 16.2.9.6 | Listing of Neurological Questionnaire Findings | L NE2 PG |
| 16.2.9.7 | Listing of Ophthalmological Examination Data | L NE1 PG |

Complete listings of all data collected in this study will also be produced.
Sponsor code: DNDI-EMO-001 Part 2

# 17.2 Data Display Specifications

#### 17.2.1 Table Outlines

#### Template T\_SD1

Table 10.1 Summary of Subject Disposition

| Population | Status | Reason for Withdrawal | Treatment 1 | Treatment 2 | Etc | All Subjects |
|---|---|---|---|---|---|---|
| Safety Population | Randomised | | | | | |
| | Completed | | | | | |
| | Withdrawn | | | | | |
| | | Death | | | | |
| | | Adverse Events | | | | |
| | | Withdrawal by subject | | | | |
| | | Physician decision | | | | |
| | | Protocol violation | | | | |
| | | Study terminated by | | | | |
| | | Sponsor | | | | |
| | | Lost to follow-up | | | | |
| | | Other | | | | |
| PK Concentration | Included | | | | | |
| PK Parameter | Included | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and column for "All emodepside"

This table will contain one column for placebo, each dose/formulation, all active and all subjects.

### Template T\_DM1

Table 14.1 Summary of Demographic Characteristics

| Variable | Statistics | Treatment 1<br>(N=xx) | Treatment 2<br>(N=xx) | Etc | All Subjects (N=xx) |
|---|---|---|---|---|---|
| Age (y) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |
| Sex | N | | | | |
| | Male | | | | |
| Race | American Indian or Alaskan | | | | |
| | Native | | | | |
| | Asian | | | | |
| | Black | | | | |
| | Native Hawaiian or other | | | | |
| | Pacific Islander | | | | |
| | White | | | | |
| | Other | | | | |
| Ethnicity | Hispanic or Latino | | | | |
| | Not Hispanic or Latino | | | | |
| Height (cm) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |
| Weight (kg) | n | | | | |
| | Mean | | | | |
| | SD | | | | |

| Variable | Statistics | Treatment 1 | Treatment 2 | Etc | All Subjects (N=xx) |
|---|---|---|---|---|---|
| | | (N=xx) | (N=xx) | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |
| BMI (kg/m2) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |
| Cigarettes* | n | | | | |
| (daily) | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |
| Alcohol* | n | | | | |
| (units/week) | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |

\*includes only those subjects who drink alcohol or smoke Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and additional demographic characteristics

#### Template T\_AE1

Table 14.3.3.xx Summary of Treatment-Emergent Adverse Events

| | | Treatme | nt 1 (N=xx) | Treatm | ent 2 (N=xx) | Etc |
|---|---|---|---|---|---|---|
| System Organ Class | Preferred Term | n | % | n | % | |
| Number of subjects with AEs | | | | | | |
| Gastrointestinal disorders | Total number of subjects | | | | | |
| | Abdominal discomfort | | | | | |
| | Abdominal pain | | | | | |
| | <b>↓</b> | | | | | |
| Nervous system disorders | Total number of subjects | | | | | |
| | Dizziness | | | | | |
| | Headache | | | | | |
| | <b>\</b> | | | | | |
| $\downarrow$ | $\downarrow$ | | | | | |

<sup>\*</sup>Subjects with ≥1 adverse event are counted only once per system organ class and preferred term.

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

SOCs and PTs are sorted in decreasing order of frequency

Presented for all applicable MedDRA system organ classes and terms. For tables by severity a sub-heading will be added to each table page

Sponsor code: DNDI-EMO-001 Part 2

#### Template T\_LB1

Table 14.3.4.xx Summary of Laboratory Values of Potential Clinical Importance

| | | Planned Relative | | Doubl | e Flags |
|----------|--------------------|------------------|---|-------|---------|
| Lab Test | Treatment | Time | n | HI | LD |
| | Treatment 1 (N=xx) | | | | |

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Source: Listing 16.2.xx

Programming notes: Continued with all tests, treatment groups and time points

#### Template T\_LB2

Table 14.3.3.2 Summary of Chemistry Laboratory Values

| - | | | | | | | | | - | Cha | ange fr | rom Baselin | ie | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned | | | | | | | | | | | | | |
| Laboratory Test (units) | Treatment | Relative Time | n | Mean | 95% CI | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| | Treatment 1 (N=xx) | -20h | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all treatments and time points.

For the summary of neurological questionnaires the first column will be headed "Questionnaire (Total Score)" and the footnote will be removed

Sponsor code: DNDI-EMO-001 Part 2

#### Template T\_UR1

Table 14.3.3.4 Summary of Urinalysis Dipstick Results

| Planned Relative | | Treatm | ent 1 (N=xx) | Treatmo | ent 2 (N=xx) |
|---|---|---|---|---|---|
| Time | Result | n | % | n | % |
| Time 1 | Positive | | | | |
| | Negative | | | | |
| | No Result | | | | |
| | Not Done | | | | |
| Time 2 | Positive | | | | |
| | Negative | | | | |
| | No Result | | | | |
| | Not Done | | | | |

Source: Listing 16.2.xx

Programming notes: Results recorded as received, e.g. Negative, Trace, etc; urine pH summarized as <5, 5-8, >8

Continued with all treatment groups and time points

#### Template T\_VS1

Table 14.3.4 Summary of Vital Signs

| | | | | | | | | | | ge from Bas | eline | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned | | | | | | | | | | | | |
| | Treatment | Relative Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Systolic BP (mmHg) | Treatment 1 (N=xx) | -20h | | | | | | | | | | | | |

Source: Listing 16.2.xx

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all variables, treatments and time points.

### Template T\_VS2

Table 14.3.4 Summary of AUCO-24 for Change from Baseline in Supine Diastolic Blood Pressure (h\*mmHg)

| | Day -1 | | | | | Day 0 | | | | Day 0 - Day -1 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | Mean | SD | Min | Max | n | Mean | SD | Min | Max | N | Mean | SD | 95% CI (Lower, Upper) |
| Treatment 1 (N=xx) | | | | | | | | | | | | | V | |

Source: Listing 16.2.xx

Difference is change from mean baseline

Programming notes: Continued with all treatments

#### Template T\_EG2

Table 14.3.5.1 Summary of ECG Values

| | | | | | | | | | Char | ige from B | aseline | 9 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned Relative | | | | | | | | | | | | |
| Variable | Treatment | Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Heart Rate (bpm) | Treatment 1 (N=xx) | -20h | | | | | | | | | | | | |
| | | -21h | | | | | | | | | | | | |
| | | -23h | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | -20h | | | | | | | | | | | | |
| | | -21h | | | | | | | | | | | | |
| | | -23h | | | | | | | | | | | | |
| PR Interval (msec) | Treatment 1 (N=xx) | -20h | | | | | | | | | | | | |
| | | -21h | | | | | | | | | | | | |
| | | -23h | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | -20h | | | | | | | | | | | | |
| | | -21h | | | | | | | | | | | | |
| | | -23h | | | | | | | | | | | | |

Sponsor code: DNDI-EMO-001 Part 2

Source: Listing 16.2.xx

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all treatment groups and time points. Do not summarise RR or QRS axis

#### Template T\_EG3

Table 14.3.7.xx Summary of ECG Values and Changes in ECG Values of Potential Clinical Importance

| | | Planned<br>Relative | 451 – 48 | 30 msec | 481, – 500 n | isec > 50 | 00 msec | 31-60<br>Increa | | >60 m | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Treatment | Time | n | % | n n | n | % | n | % | n | % |
| QT interval | Treatment 1 | 1h | | | | | | | | | |
| | (N=xx) | 2h | | | | | | | | | |
| | | 3h | | | | | | | | | |
| | Treatment 2 | 1h | | | | | | | | | |
| | (N=xx) | 2h | | | | | | | | | |
| | | 3h | | | | | | | | | |
| QTcB interval | Treatment 1 | 1h | | | | | | | | | |
| | (N=xx) | 2h | | | | | | | | | |
| | | 3h | | | | | | | | | |
| | Treatment 2 | 1h | | | | | | | | | |
| | (N=xx) | 2h | | | | | | | | | |
| | | 3h | | | | | | | | | |

Source: Listing 16.2.xx

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all treatments, variables and time points.

#### Template T\_PE1

Table 14.3.8.xx Summary of Physical Examination Data

| | Planned | | | |
|--------------------|----------|--------------|-------------|-------------|
| | Relative | | Treatment 1 | Treatment 2 |
| Body System | Time | Result | (N=xx) | (N=xx) |
| General Appearance | Time 1 | Normal | n (%) | |
| | | Abnormal NCS | x (xx) | |
| | | Abnormal CS | | |
| | Time 2 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |
| HEENT | Time 1 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |
| | Time 2 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |

Source: Listing 16.2.xx

Programming notes: Continued with all body system, treatments and time points. Include rows for each outcome in CRF

If results are missing "missing" row will be added. Percentages calculated using the number of available results as denominator.

Template T\_NE1

Table 14.3.8.xx Summary of Neurological Examination Data

Mental Status

| | Planned | | | |
|-------------|----------|--------------|-------------|-------------|
| | Relative | | Treatment 1 | Treatment 2 |
| Body System | Time | Result | (N=xx) | (N=xx) |
| | | | n (%) | n (%) |
| Alertness | Time 1 | Normal | x (xx) | |
| | | Abnormal NCS | x (xx) | |
| | | Abnormal CS | | |
| | Time 2 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |
| Speech | Time 1 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |
| | Time 2 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |

Source: Listing 16.2.xx

Programming notes: Continued with all examinations/test, treatments and time points. Include rows for each outcome in CRF

For Ophthalmological assessment, replace body system with Test

If results are missing "missing" row will be added. Percentages calculated using the number of available results as denominator.

 ${\it Use PESCAT as subheading (not for Ophthalmological Assessment)}.$ 

Sponsor code: DNDI-EMO-001 Part 2

#### Template T\_PK1

Table 14..2.xx Summary of Emodepside Plasma Pharmacokinetic Concentration-Time Data [units]

| | | Planned<br>Relative | | No. | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | N | Time | n | Imputed | Mean | 95% CI | SD | %CV | Median | Min | Max |
| Dose 1 | | 1h | | | | | | | | | |
| Dose 2 | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and timepoints

Means, SD, CI and CV should only be calculated if ≥2/3 individual values are >LLOQ

#### Template T\_PK3

Table 14..2.xx Summary of Derived Emodepside Plasma Pharmacokinetic Parameters

| Parameter | Treatment | N n | Mean | 95% CI | SD | %CV | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|
| AUC <sub>last</sub> (units)<br>C <sub>max</sub> (units) | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and parameters

Sponsor code: DNDI-EMO-001 Part 2

#### Template T\_PK4

Table 14..2.xx Summary of Log-Transformed Derived Emodepside Plasma Pharmacokinetic Parameters

| Parameter | Treatment | N | n | Geom Mean | 95% CI | SD (logs) {%CVb} |
|---|---|---|---|---|---|---|
| AUC <sub>last</sub> (units)<br>C <sub>max</sub> (units) | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and parameters

#### Template T\_PK7

Table 14.2.xx Assessment of the Effects of Food on the PK of Emodepside

| | | | LS Means | | |
|---|---|---|---|---|---|
| Parameter | Treatment | Fed | Fasted | Ratio | 90% CI |
| | | | | (Fed/Fasted) | |
| Cmax (Units) | | xxxx.xx | XXXX.XX | xxxx.xx | (xxxx.xx, xxxx.xx) |

Source: Listing 16.2.xx

Programming notes: Continued with AUC<sub>inf</sub>,

Sponsor code: DNDI-EMO-001 Part 2

#### Template T\_PD1

Table 14...xx Summary of Glucose

| | | | | | | | | | | Ch | ange f | rom Baselin | e | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | | | | | | | | | | | | | |
| Treatment | Relative Time | n | Mean | 95% CI | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Treatment 1 (N=xx) | -24h | х | x | x | х | x | х | х | | | | | | |
| | -20h | х | x | х | х | х | х | x | x | х | x | x | Х | X |

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all PD parameters, treatments and timepoints

Change from baseline calculated from "pre-dose" on each day

### Template T\_PD2

Table 14...xx Summary of Difference Between Day -1 and Day 0 in Glucose

| | Planned Relative Time | Relative Time Day -1 – Day 0 | | | |
|---|---|---|---|---|---|
| Treatment | | n | Mean | SD | 95% CI |
| Treatment 1 (N=xx) | | | | | |

Note: Difference is change from baseline

Programming notes: Continued with time points and treatments

Sponsor code: DNDI-EMO-001 Part 2

## Template T\_PD3

Table 14...xx Summary of AUC<sub>0-24</sub> for change from baseline in Glucose (units)

| | Day -1 | | | | Day 0 | | | | Day -1 – Day 0 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | Mean | SD | Min | Max | n | Mean | SD | Min | Max | n | Mean | SD | 95% CI |
| Treatment 1 (N=xx) | | | | | | | | | | | | | | |

Note: Difference is change from baseline

Programming notes: Continued with all treatments

## 17.2.2 Figure Outlines

#### Template F\_PK1

Figure 16.2.4 .xx Individual Emodepside Plasma Concentration-Time Plots (Linear and Semi-log)



Programming note: Plot will include all subjects for a given treatment group

#### Template F\_PK2

Figure 16.2.4.xx Geometric mean (+ SD) of Emodepside Plasma Concentration-Time Plots (Linear and Semi-log)





Programming note: The SD is the geometric standard deviations

#### Template F\_PK10

Figure 16.2.xx Individual Emodepside Plasma Concentration-Time Plots (log scale) for Estimation of Lambda-z, with Regression Line



#### Template F\_PD1

Figure **16.2.**xx Individual Glucose-Time Plots



Programming note: Continue with Insulin, Glucagon and Cortisol land normal rages as reference lines.

For Blood pressure and Heart Rate, include PCI limits as reference lines.

Plot will include all subjects for a given treatment group

4 plots per page

### Template F\_PD2

Figure 16.2.xx Individual Glucose and PK Concentration Plots - Including Related Significantly Important AE Durations



Cohorts with at least 1 related significant AE displayed

Programming note: Continue with Insulin
2 plots per page

Sponsor code: DNDI-EMO-001 Part 2

## 17.2.3 Listing Outlines

#### Template L\_SD1\_PG

Listing 16.2.x.xx Listing of Study Dates

Treatment Subject Screening Day -1 Day 0 Follow-Up

Programming notes: Lists dates for screening, each dosing period and follow up

#### Template L\_SD2\_PG

Listing 16.2.x.xx Listing of Reasons for Withdrawal

Date of Study

Treatment Subject Withdrawal Day Reason

#### Template L\_DV1\_PG

Listing of Subjects with Inclusion/Exclusion Criteria Deviations Listing 16.2.x.xx

Treatment Subject Type Criterion Inclusion

Exclusion

Sponsor code: DNDI-EMO-001 Part 2

Template L\_TD1\_PG

Listing 16.2.x.xx Listing of Subjects with Time Deviations

Allowed Actual deviation deviati

Only include time deviations which exceed the allowed deviation

deviation deviation

Procedure (h:min) (h:min)

Template L\_DV2\_PG

**Programming notes:** 

Treatment

Subject

Listing 16.2.2.3 Listing of Subjects with Other Protocol Deviations

Timepoint

Treatment Subject Protocol Deviation

Template L\_AN1\_PG

Listing 16.2.x.xx Listing of Analysis Populations

Treatment Subject Safety Population PK concentration

Programming notes: continue for all populations

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_DM1\_PG

Listing 16.2.x.xx Listing of Demographic Characteristics

| | | | | | | | | | | | Alcohol | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Height | Weight | | Consumption | Cigarettes |
| Treatment | Subject | Date of visit | Date of birth | Age (y) | Gender | Race | Ethnicity | (cm) | (kg) | BMI (kg/m2) | (units/week) | (daily) |

Treatment 1



#### Template L\_CM1\_PG

Listing 16.2.x.xx Listing of Concomitant Medications

| | | | Dose/ | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Drug Name/ | Units/ Freq/ | Date/time Started/ | Time Since Last | Started | Pre- | Ongoing |
| Treatment | Subject | Indication | Route | Date Stopped | Dose | Trial? | | Medication? |

#### Template L\_EX1\_PG

Listing 16.2.x.xx Listing of Exposure Data

| | | | | Dur- | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Start Date/ | Stop Date/ | ation | | Dose | Formulation | n/ |
| Treatment | Subject | Start Time of Dose | Stop Time of Dose | (days) | Dose | Unit | Route | Frequency |
| Treatment 1 | 1001 | 01JAN2002/ | 15FEB2002/ | 46 | 25 | mg | Tablet/ | 2xday |
| | | 23:59 | 15:30 | | | | Oral | |

## Template L\_AE1\_PG

Listing 16.2.x.xx Listing of All Adverse Events

| | | | | | | Frequency/ Action | Related to Study |
|---|---|---|---|---|---|---|---|
| | | SYSTEM ORGAN CLASS/ | Outcome/ Onset | | Severity/ | Taken (1)/ | Drug/ |
| | | PREFERRED TERM/ | Date/Time/ Resolved | Time Since Last | Serious/ | Other Action | Treatment |
| Treatment | Subject | Verbatim Text | Date/Time/ Duration | Dose | Withdrawal | Taken | Emergent? |
| Treatment 1 | 1001 | GASTROINTESTINAL | Resolved/ | 10d 7h 3m | Mild/ | Intermittent/ Dose | Possibly/ |
| | | DISORDERS / | 24SEP2003/13:05/ | | No/ | not changed/ | Yes |
| | | INTESTINAL SPASM/ | 27OCT2003/7:50/ | | Yes | None | |
| | | Entero-spasm | 34d 4h 5m | | | | |

<sup>(1)</sup> Action Taken with Study Treatment

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_LB1\_PG

Listing 16.2.x.xx Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance

| | | | Planned<br>Relative | | Study | | | | | Clinically |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Laboratory test (units) | Time | Date/Time | Day | Value | Normal Range | NR | BL | Significant? |
| Treatment 1 | 1001 | Alk Phos (U/L) | Time 1 | 01JAN2002/ | -1 | 64.00 | 32.0- 92.0 | | | |
| | | | | 13:34 | | | | | | |
| | | | Time 2 | 01APR2002/ | 85 | 84.00 | 32.0- 92.0 | | | |
| | | | | 07:22 | | | | | | |
| | | ALT (U/L) | Time 1 | 01JAN2002/ | -1 | 29.00 | 10.0- 40.0 | | | |
| | | | | 18:56 | | | | | | |
| | | | Time 2 | 01APR2002/ | 85 | 70.00 | 10.0- 40.0 | Н | - 1 | Υ |
| | | | | 09:22 | | | | | | |

NR for Normal Range flag, BL for Change from Baseline flag;

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Programming notes: Lists only double-flagged subjects

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_LB2\_PG

Listing 16.2.x.xx Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities

| | | Planned<br>Relative | | Alkaline | Phosphata | se (IU/L) | Alanine | Amino Tra<br>(IU/L) | nsferase | Aspartate | Amino Tran | sferase | Total B | Silirubin (UN | MOL/L) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Time | Date/Time | Result | NR | BL | Result | NR | BL | Result | NR | BL | Result | NR ` | BL |
| | | Planned | | | | | | | | | | | | | |
| | | Relative | | Chlo | ride (MMC | DL/L) | Gluc | ose (MMC | L/L) | Potas | sium (MMOL | L/L) | Sod | ium (MMO | L/L) |
| Treatment | Subject | Time | Date/Time | Result | NR | BL | Result | NR | BL | Result | NR | BL | Result | NR | BL |
| | | | Planned | | | | | | | | | | | | |
| | | | Relative | | | Calcium | (MMOL/L) | | Creatinin | ie (UMOL/L) | | | Etc. | | |

NR for Normal Range flag, BL for Change from Baseline flag;

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Programming notes: Lists only double-flagged subjects

*Include all parameters for the study following the order from the lab report (above is a guide only)* 

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_URI

Listing 16.2.x.xx Listing of Urinalysis Data

| | | Planned | | Specific | Gravity | рН | ł | Prot | ein | Gluc | cose |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Relative | | | | | | | | | |
| Treatment | Subject | Time | Date/Time | Result | NR | Result | NR | Result | NR | Result | NR |

NR for Reference interval flag, H = Above reference interval, L = Below reference interval

Programming notes: Include all parameters for the study following the order from the lab report (above is a guide only)

#### Template L\_VS1\_PG

Listing 16.2.x.xx Listing of Vital Signs of Potential Clinical Importance

| | | | | Systolic | Diastolic | |
|---|---|---|---|---|---|---|
| | | Planned Relative | | Blood Pressure | Blood Pressure | Etc |
| Treatment | Subject | Time | Date/Time | (mmHg) | (mmHg) | (units) |
| | | 24 H | 26SEP2012:09:57 | 63 | 148* | |

<sup>\*</sup> Value of potential clinical importance

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_EG1\_PG

Listing 16.2.x.xx Listing of ECG Values of Potential Clinical Importance

| | | | | | | | QT Int | . (msec) | QTcB | (msec) | QTcF | (msec) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Subject | Planned<br>Relative Time | Date/Time | Heart<br>Rate<br>(bpm) | PR Int.<br>(msec) | QRS<br>Dur.<br>(msec) | QRS<br>Axis<br>(deg) | Observed | Change<br>from<br>Baseline | Observed | Change<br>from<br>Baseline | Observed | Change<br>from<br>Baseline |
| | Pre-dose (1) | 26SEP2012:09:57 | 63 | 148 | 78 | 50 | 390 | 32.7 * | 399 | -27.7 | 419 | -11 |
| | Pre-dose (2) | | | | | | | | | | | |
| | Pre-dose (3) | | | | | | | | | | | |
| | Mean Pre-dose | | | | | | | | | | | |
| | 24 H | | | | | | | | | | | |

<sup>\*</sup> Value of potential clinical importance

Programming notes: Do not list RR

#### Template L\_EG2\_PG

Listing 16.2.x.xx Listing of Abnormal ECG Findings

| | | | | | Comment on |
|---|---|---|---|---|---|
| | | Planned Relative | | | Clinical |
| Treatment | Subject | Time | Date/Time | ECG Finding | Significance |

Programming notes: Lists only values with Normal variant='No' or with comment on ECG result

ECG Finding contains Physician's Opinion from CRF and relates to whole trace (not individual parameters), e.g. Normal, Abnormal - NCS or Abnormal - CS

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_PE1\_PG

Listing 16.2.x.xx Listing of Abnormal Physical Examination Findings

Planned Relative

Treatment Subject Time Date/Time Site Details

Programming Notes: List only findings with an 'Abnormal NCS' or 'Abnormal CS' result.

If subjects have multiple abnormal sites at a given time, create a separate row for each site.

#### Template L\_NE1\_PG

Listing 16.2.x.xx Listing of Neurological Examination Findings

Planned

Treatment Subject Relative Time Date/Time Type Assessment Details

Programming Notes: Type = (Mental Status, Mood, Cranial Nerves etc.

List all findings

If subjects have multiple abnormal assessment at a given time, create a separate row for each assessment.

For Ophthalmological assessment, the columns will be Treatment, Subject, Planned relative Time, Date/Time, Test and Details

#### Template L\_NE2\_PG

Listing 16.2.x.xx Listing of Neurological Questionnaire Findings

Mental Status

Total Score
Hamilton Epworth

Planned Relative Depression Sleepiness

Treatment Subject Time Date/Time Rating Scale Score BDI-II

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_PK1\_PG

Treatment

Listing 16.2.4.xx Listing of Emodepside Plasma Pharmacokinetic Con centration-Time Data

{Add. time

var.}

Planned Study Day **Relative Time** Date

Time Deviation Actual Relative (units)

Time

Concentration (units)

BLQ = Below Limit of Quantification

Programming notes: Values below LLOQ are shown as BLQ

For PD: BLQ values are imputed to half LLOQ

For the listings of derived AUCO-24 PD concentrations, the columns will be Treatment, Subject, Planned Relative Time, Concentrations (units)

#### Template L\_PK3\_PG

Listing 16.2.4 xx Listing of Emodepside Urine Excretion Rate Data

Planned

Relative

Urine Conc.

Treatment

Subject

Subject

Time

Stop Date/Time Start Date/Time

(units)

Total Sample Volume (mL)

Actual time

Amount excreted (units)

#### Template L\_PK4\_PG

Listing 16.2.4.xx Listing of Derived Emodepside Pharmacokinetic Parameters

{Add.

time Treatment Subject var.}

AUCinf (units)

AUC<sub>t</sub> (units)

 $C_{\mathsf{max}}$ (units)

 $t_{1/2}$ (units)

 $t_{\mathsf{max}}$ (units)

Programming notes:

Continue with all parameters

# **Appendix A: Laboratory Ranges**

## Pre-determined Changes for Laboratory Data (from FL140 v3)

| | | | | Delta | ranges |
|---|---|---|---|---|---|
| Test | Test Code | Unit | Sex | Acceptable decrease | Acceptable increase |
| Activated partial thromboplastin time | APTTT | sec | Both | - 8.0 | + 8.0 |
| Alanine transferase | ALTN | IU/L | F | - | + 30 |
| Alanine transferase | ALTN | IU/L | M | _ | + 30 |
| Albumin | ALB | g/L | Both | - 7.5 | + 7.5 |
| Alkaline phosphatase | ALPN | IU/L | Both | - 30 | + 30 |
| Amylase | AMY | U/L | Both | - | + 150 |
| Aspartate transferase | ASTN | IU/L | F | - 30 | + 30 |
| Aspartate transferase | ASTN | IU/L | M | - 30 | + 30 |
| Basophils | BASO | 10 <sup>9</sup> /L | Both | - | + 0.3 |
| Bilirubin conjugated | DBIL | μmol/L | Both | - | + 4.0 |
| Bilirubin total | TBIL | μmol/L | F | - 20 | + 10.0 |
| Bilirubin total | TBIL | μmol/L | M | - 20 | + 10.0 |
| Bilirubin unconjugated | IBIL | μmol/L | Both | - | - |
| C-reactive protein | CRP | mg/L | Both | - | - |
| CK relative index | CKMBR | % | Both | - | _ |
| Calcium | CA | mmol/L | Both | - 0.4 | + 0.4 |
| Carbon dioxide | CO2 | mmol/L | Both | - 8 | + 8 |
| Chloride | CL | mmol/L | Both | - 10 | + 10 |
| Cholesterol | CHOL | mmol/L | Both | - | + 0.7 |
| Creatine kinase | CK | IU/L | F | - | + 400 |
| Creatine kinase | CK | IU/L | M | - | + 400 |
| Creatinine | CREA | μmol/L | Both | - | + 40 |
| Creatinine (DOA urine) | CREDA-U | mmol/L | Both | - | - |
| Eosinophils | EOS | 10 <sup>9</sup> /L | Both | - | + 0.5 |
| Erythrocyte sedimentation rate | ESR | mm/h | Both | - | - |
| Fibrinogen | FIB-C | g/L | Both | - | - |
| Free T3 | FT3 | pmol/L | Both | - 3.5 | + 3.5 |
| Free T4 | FT4 | pmol/L | Both | - 15 | + 15 |
| Gamma glutamyl transferase | GGT | IU/L | F | - | + 40 |
| Gamma glutamyl transferase | GGT | IU/L | M | - | + 40 |
| Globulin | GLOB | g/L | Both | - 7.5 | - |
| Glucose | GLU | mmol/L | Both | - 1.5 | + 2.5 |
| Haematocrit | HCT | L/L | Both | - 0.05 | - |
| Haemoglobin | HB | g/L | Both | - 20 | - |
| High density lipoprotein | HDL | mmol/L | Both | - 1.5 | + 1.5 |
| International normalised ratio | INRR | ratio | Both | - | - |
| Lactate dehydrogenase | LDH | IU/L | Both | - | + 150 |
| Lymphocytes | LYMP | 10 <sup>9</sup> /L | Both | - 1.5 | + 1.5 |
| Magnesium | MG | mmol/L | Both | - | - |
| Mean cell haemoglobin | MCH | pg | Both | - 2 | + 2 |
| Mean cell haemoglobin concentration | MCHC | g/L | Both | - 25 | + 25 |
| Mean cell volume | MCV | fL | Both | - 10 | + 10 |

| | | | | Delta ranges | |
|---|---|---|---|---|---|
| Test | Test Code | Unit | Sex | Acceptable decrease | Acceptable increase |
| Monocytes | MONO | 10 <sup>9</sup> /L | Both | - 0.50 | + 0.5 |
| Neutrophils | NEUT | 10 <sup>9</sup> /L | Both | - 2 | + 8 |
| Phosphate | PHOS | mmol/L | Both | - 1 | + 1 |
| Platelets | PLT | 10 <sup>9</sup> /L | Both | - 100 | + 100 |
| Platelets (citrate tube) | PLTC | 10 <sup>9</sup> /L | Both | - 100 | + 100 |
| Potassium | K | mmol/L | Both | - 0.75 | + 0.75 |
| Prolactin | PROL | μg/L | Both | - | - |
| Prothrombin time | PTT | sec | Both | -4.0 | + 4.0 |
| Red blood cells | RBC | $10^{12}/L$ | Both | - 1.0 | - |
| Reticulocyte | RET | % | Both | - | - |
| Reticulocyte count | RETC | 10 <sup>9</sup> /L | Both | - | - |
| Reticulocyte manual count | RETM | 10 <sup>9</sup> /L | Both | - | - |
| Sodium | NA | mmol/L | Both | - 8 | + 8 |
| Thrombin time | TT | sec | Both | - | - |
| Thyroid stimulating hormone | TSH | mIU/L | Both | - 3 | + 3 |
| Total protein | TP | g/L | Both | - 15 | - |
| Triglycerides | TG | mmol/L | Both | - | + 1.5 |
| Urea | UREA | mmol/L | Both | - 5 | + 2 |
| Uric acid | UA | μmol/L | Both | - 100 | + 100 |
| Urine pH | UPH | N/A | Both | - 4 | + 4 |
| Urine red blood cells | URBC | $10^{6}/L$ | Both | - | + 10 |
| Urine white blood cells | UWBC | $10^{6}/L$ | Both | - | + 100 |
| White blood cells | WBC | 10 <sup>9</sup> /L | Both | - 2 | + 8 |

## **Appendix B: Pharmacokinetic Analysis**

### 1 Calculation Methods

## 1.1 Data Handling Conventions

#### 1.1.1 Actual v Planned Times

Actual sample times will be used for the calculation of pharmacokinetic parameters and for individual concentration-time plots.

Planned sampling times will be used to calculate the concentration-time summary statistics and summary concentration-time plots.

### 1.1.2 Missing and BQL Concentrations

Missing values will not be used in any way.

For calculation of all pharmacokinetic parameters and individual profile plots, plasma concentrations below the quantifiable limit (BQL) of the assay will not be used for the calculation of PK parameters (except BQL values observed at time points before the maximum concentration, which will be taken as zero).

BQL values will be substituted by one half of the lower limit of quantification for calculation of plasma concentration summary statistics. The number of imputed values will be included in the summary table.

For urine concentrations reported as BQL it is not possible to impute a value. The amount excreted will be set to zero when concentration is BQL.

#### 1.2 AUC Calculations

The AUC will be calculated by a combination of linear and logarithmic methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations

 $AUC_{(0-\infty)}$  values with <20% of this area extrapolated will be reported.

Sponsor code: DNDI-EMO-001 Part 2

It is acceptable to include data from profiles with >20% extrapolated as long as at least 80% of the profiles in the study have <20% of the  $AUC_{(0-\infty)}$  as extrapolated area. In this instance, individual plasma concentration-time profiles for which the extrapolated areas are >20% of  $AUC_{(0-\infty)}$  will be identified.

It is unacceptable to use  $AUC_{(0-\infty)}$  data if >40% of the AUC has been extrapolated, except in specific situations which should be carefully justified in the study report.

#### 1.3 Lambda-z Calculations

The apparent terminal phase rate-constant ( $\lambda_z$ ) will be estimated by linear regression of logarithmically transformed concentration versus time data. Only those data points which are judged to describe the terminal log-linear decline will be used in the regression.

During the analysis, repeated regressions are carried out using the last three points with non-zero concentrations, then the last four points, last five, etc. Points prior to  $C_{max}$  are not used. Points with a value of zero for the concentration are excluded. For each regression, an adjusted  $R^2$  is computed. The  $\lambda_z$  using the regression with the largest adjusted  $R^2$  is selected. If the adjusted  $R^2$  does not improve, but is within 0.0001 of the largest adjusted  $R^2$  value, the regression with the larger number of points is used.  $\lambda_z$  must be positive, and calculated from at least three data points.

For non-compartmental analysis uniform weighting will be applied.

#### 1.4 Observed v Predicted Values

For parameters dependent on  $\lambda_z$ , the 'predicted' rather than the 'observed' parameters will be calculated.

The 'predicted' parameters are calculated using  $\hat{C}_t$  (the predicted value of the concentration at time tn); whilst the 'observed' parameters use the last observed concentration.

## 2 General Considerations for Data Analysis

### 2.1 Derived and transformed data

In general, concentration and concentration-related quantities, rate constants and half-lives (e.g.  $C_{max}$ , AUC,  $t_{1/2}$ , CL/F,  $V_z$ /F and MRT) will be analysed after logarithmic transformation. Logarithmic transformations will use natural logarithms (log<sub>e</sub>). A list of those parameters that will be log transformed are given below.

## 2.2 Summary data

Means at any time will only be calculated if at least 2/3 of the individual data are measured and are above the lower of quantification (LLOQ).

# 3 Parameter Definitions

## 3.1 Plasma Parameters

# 3.1.1 Emodepside

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| Concentrations and | | | | | | | |
| C <sub>max</sub> | Maximum (peak) plasma concentration | The maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | ng/mL | Y | Cmax | CMAX | $C_{max}$ |
| C <sub>max</sub> /D | Dose-normalised C <sub>max</sub> to infinity | The dose-normalised $C_{max}$ will be calculated as $C_{max}$ /Dose administered | (ng/mL)/mg | Y | Cmax_D | CMAXD | C <sub>max</sub> /D |
| $C_{max,norm}$ | Observed maximum plasma concentration corrected by dose and body weight | The C <sub>max</sub> normalised by dose and body weight will be calculated as C <sub>max</sub> /(Dose administered*body weight) | (ng/mL)/(mg*kg) | Y | N/A | CMAXWD | $C_{\text{max,norm}}$ |
| t <sub>max</sub> | Time to reach maximum (peak) plasma concentration | The first time of maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | h | N | Tmax | TMAX | t <sub>max</sub> |
| Half-life | | | | | | | |
| $\lambda_z$ | Terminal rate constant | The apparent terminal phase rate-constant $(\lambda_z)$ will be estimated by linear regression of logarithmically transformed concentration versus time data. | 1/h | Y | Lambda_z | LAMZ | $\lambda_{\mathrm{z}}$ |
| Point terminal | Number of points for<br>Lambda z | The number of time points used in calculating Lambda z | - | - | No_points_lambda<br>_z | LAMZNPT | $n_{ m pts}$ |
| t <sub>½</sub> | Terminal half-life | The terminal half-life calculated from the terminal slope of the log concentration-time curve, as follows: $t_{1/2} = \frac{\log_e 2}{\lambda_z}$ | h | Y | HL_Lambda_z | LAMZHL | t <sub>1/2</sub> |
| t <sub>½,0-24</sub> | Dominant half-life | The half-life calculated from the terminal slope of the log concentration-time (0-24h) curve, as follows: $t_{1/2} = \frac{\log_e 2}{\lambda_z}$ | h | Y | HL_Lambda_z | TBC | t <sub>1/2,0-24</sub> |

Sponsor code: DNDI-EMO-001 Part 2

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| Areas under the cur | rve | | | | | | |
| AUCt | Area under the plasma<br>concentration-time curve<br>from time zero to time of last<br>measurable concentration | The area under the concentration-time curve from zero time (pre-dose) to the time of last quantifiable concentration will be calculated using the (specified) trapezoidal method. | h*ng/mL | Y | AUClast | AUCLST | AUC <sub>last</sub> |
| $\mathrm{AUC}_{\mathrm{t,norm}}$ | Area under the concentration-time curve from time zero (pre-dose) to the time of last quantifiable concentration corrected by dose and body weight | The AUC normalised by dose and body weight will be calculated as AUC <sub>t</sub> /(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | N/A | AUCLSTWD | AUC <sub>last,norm</sub> |
| AUC <sub>1-∞</sub> | Area under the exponential curve from t <sub>last</sub> to infinity | The area under the exponential curve from $t_{last}$ to infinity, calculated as follows: $AUC_{t-\infty} = \frac{\hat{C}_t}{\lambda_z} \text{ where } \hat{C}_t \text{ is the }$ predicted value of the concentration at $t_{last}$ . | h*ng/mL | N/A | N/A | AUCIFO | AUCt-inf |
| $\mathrm{AUC}_{\infty}$ | Area under the plasma concentration-time curve from time zero to infinity | The area under the concentration-time curve will be calculated using the (specified) trapezoidal method for the interval 0 to $t_{last}$ (time $t_{last}$ is the time at which the last non-zero level was recorded), plus $AUC_{t-\infty}$ . | h*ng/mL | Y | AUCINF_pred | AUCIFP | $\mathrm{AUC}_{\mathrm{inf}}$ |
| AUC∞/Dose | Dose-normalised AUC to infinity | The dose-normalised AUC to infinity will be calculated as AUC <sub>∞</sub> /Dose administered | (h*ng/mL)/mg | Y | AUCINF_D_pred | AUCIFPD | AUC <sub>inf</sub> /D |
| $\mathrm{AUC}_{\infty,\mathrm{norm}}$ | Area under the concentration-time curve from time zero to infinity corrected by dose and body weight | The AUC normalised by dose and body weight will be calculated as AUC <sub>x</sub> /(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | N/A | AUCIFPWD | AUC <sub>inf,norm</sub> |
| %AUC <sub>extrap</sub> | Percentage of $AUC_{\infty}$ extrapolated from from $t_{last}$ to infinity | $\% AUC_{extrap} = \frac{100 \times AUC_{t-\infty}}{AUC_{\infty}}$ | % | N | AUC_%EXTRAP<br>_pred | AUCPEP | %AUC <sub>extrap</sub> |
| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| AUC <sub>0-24</sub> | Area under the plasma concentration-time curve from time zero to 24h | The area under the concentration-time curve from zero time (pre-dose) to 24h will be calculated using the (specified) trapezoidal method. If $\lambda_z$ is not estimable, a partial AUC is not calculated (when $t_{last} < t$ ). | h*ng/mL | Y | User specified area | AUCINT | AUC <sub>24</sub> |
| AUC <sub>0-24</sub> /D | Dose-normalised AUC from time zero to 24h | The dose-normalised AUC from time zero to 24h will be calculated as AUC <sub>0-24</sub> /Dose administered | (h*ng/mL)/mg | Y | N/A | AUCINTD | AUC <sub>24</sub> /D |
| AUC <sub>0-24,norm</sub> | Area under the concentration-time curve from time zero to 24h corrected by dose and body weight | The AUC from time zero to 24h normalised by dose and body weight will be calculated as AUC <sub>0-24</sub> /(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | N/A | AUCINTWD | AUClast,norm |
| | of distribution and mean residen | | | | | | |
| CL/F | Apparent total clearance from plasma after oral administration | Apparent total clearance from plasma will be calculated using the following formula: $CL/F = \frac{Dose}{AUC_{\infty}}$ | L/h | Y | Cl_pred (actually derives Cl_F_pred for oral dose) | CLFP | CL/F |
| V <sub>z</sub> /F | Apparent volume of<br>distribution during terminal<br>phase after non-intravenous<br>administration | Apparent volume of distribution will be calculated using the following formula: $V_z / F = \frac{Dose}{\lambda_z \bullet AUC_{\infty}}$ | L | Y | Vz_pred (actually derives Vz_F_pred for oral dose) | VZFP | V <sub>z</sub> /F |
| MRT | Mean Residence Time | The mean residence time will be calculated using: $MRT = \frac{AUMC}{AUC_{\infty}}$ | h | Y | MRTINF_pred | MRTIFP | MRT |
| AUMC | Area under the first moment of the plasma concentration-time curve from time zero to infinity | The area under the first moment of the concentration-time curve from zero time (predose) extrapolated to infinite time will using the (specified) trapezoidal method, as for AUC. | h <sup>2</sup> *ng/mL | - | AUMCINF_pred | AUMCIFP | AUMC |

HMR code: 15-020 Part 2

Sponsor code: DNDI-EMO-001 Part 2

# **Appendix C: Sample Page Layout**

| DNDi: DNDI-EMO-001 | | Page x of y |
|---|---|---|
| Population: [Pop] | | |
| | Table [number] [title] | |
| | Column headers | |
| | Main body of output | |
| | Source: Listing [16.2.xx] | |
| Footnotes about the table or listing text | go here. | |
| Program: [Prog Name] | [Date] | HMR 15-020 Part 2 |
| Produced By:[Username] | | |

Font size will be Arial 9.5pt. The following margins will be used: Left: 1", Right: 1", Top: 1", Bottom: 1"

<sup>\*</sup>y = last page of individual output

# **Table of contents**

| 1 | LIST | OF ABBREVIATIONS | 5 |
|----|------|------------------------------------------------------------|----|
| 2 | SIGN | NATURES | 7 |
| 3 | INTE | RODUCTION | 8 |
| 4 | STUI | DY OBJECTIVE(S) AND ENDPOINT(S) | 8 |
| | 4.1 | Study Objective(s) | 8 |
| | | 4.1.1 Primary Objective(s) | |
| | | 4.1.2 Secondary Objective(s) | |
| | 4.2 | Study Endpoint(s) | |
| | | 4.2.1 Safety and Tolerability Variables: | |
| | | 4.2.2 Pharmacokinetic Variables: | |
| | | 4.2.3 Pharmacodynamic Variables: | |
| | 4.3 | Statistical Hypotheses | |
| 5 | STUI | DY DESIGN | 10 |
| 6 | PLA | NNED ANALYSES | 17 |
| | 6.1 | Interim Analyses | 17 |
| | | 6.1.1 Persons responsible for analysis | |
| | 6.2 | Final Analysis | 17 |
| | | 6.2.1 Persons responsible for analysis | |
| 7 | SAM | PLE SIZE CONSIDERATIONS | 17 |
| | 7.1 | Sample Size Assumptions | 17 |
| 8 | ANA | LYSIS POPULATIONS | 18 |
| | 8.1 | Analysis Datasets | 18 |
| 9 | TRE | ATMENT COMPARISONS | 18 |
| | 9.1 | Data Display Treatment and Other Subgroup Descriptors | 18 |
| | | 9.1.1 Conventions for Summary Statistics and Data Displays | 19 |
| 10 | DAT | A HANDLING CONVENTIONS | 19 |
| | 10.1 | Premature Withdrawal and Missing Data | 19 |
| | 10.2 | Derived and Transformed Data | 20 |
| | 10.3 | Assessment Windows | 20 |
| | 10.4 | Values of Potential Clinical Importance | 20 |
| 11 | STUI | DY POPULATION | 21 |
| | 11.1 | Disposition of Subjects | |
| | 11.2 | Protocol Deviations | 21 |
| | 11.3 | Demographic and Baseline Characteristics | 22 |
| | | <del>-</del> | |

| | 11.4 | Treatment Compliance | 22 |
|---|---|---|---|
| 12 | SAFE | TY ANALYSES | 22 |
| | 12.1 | Extent of Exposure | 22 |
| | 12.2 | Adverse Events | 22 |
| | 12.3 | Deaths and Serious Adverse Events | 23 |
| | 12.4 | Adverse Events Leading to Withdrawal from the Study | 23 |
| | 12.5 | Clinical Laboratory Evaluations | 23 |
| | 12.6 | Other Safety Measures | 24 |
| | | 12.6.1 Vital signs | 24 |
| | | 12.6.2 ECG | 24 |
| | | 12.6.3 Neurological examination | |
| | | 12.6.4 Physical examination | |
| | | 12.6.5 Ophthalmology assessments | |
| 13 | PHAR | RMACOKINETIC ANALYSES | |
| | 13.1 | Plasma PK | 25 |
| | | 13.1.1 Pharmacokinetic Concentration Data | |
| | | 13.1.2 Pharmacokinetic Parameters | |
| | 13.2 | Urinary PK | |
| 14 | PHAR | RMACODYNAMIC ANALYSES | 26 |
| 15 | CHAN<br>27 | NGES FROM THE PROTOCOL SPECIFIED STATISTICAL A | ANALYSIS |
| 16 | REFE | RENCES | 27 |
| 17 | ATTA | ACHMENTS | 29 |
| | 17.1 | Table of Contents for Data Display Specifications | 29 |
| | 17.2 | Data Display Specifications | 36 |
| | | 17.2.1 Table Outlines | |
| | | 17.2.2 Figure Outlines | 50 |
| | | 17.2.3 Listing Outlines | 55 |
| APPI | ENDIX | A: LABORATORY RANGES | 65 |
| APPI | ENDIX | B: PHARMACOKINETIC ANALYSIS | 67 |
| 1 | CALC | CULATION METHODS | 67 |
| | 1.1 | Data Handling Conventions | 67 |
| | | 1.1.1 Actual v Planned Times | |
| | | 1.1.2 Missing and BQL Concentrations | 67 |
| | 1.2 | AUC Calculations | 67 |
| | 1.3 | Lambda-z Calculations | 68 |
| | 1.4 | Observed v Predicted Values | 68 |

| 2 | GEN | IERAL CONSIDERATIONS FOR DATA ANALYSIS | 69 |
|-----|--------|----------------------------------------|----|
| | 2.1 | Derived and transformed data | 69 |
| | 2.2 | Summary data | 69 |
| 3 | PAR | AMETER DEFINITIONS | 70 |
| | 3.1 | Plasma Parameters | 70 |
| | | 3.1.1 Emodepside | 70 |
| ΔPI | PENDIS | X C. SAMPLE PAGE LAVOUT | 73 |

### 1 List of abbreviations

Terminal rate constant  $\lambda_z$ AΕ Adverse Event ANOVA Analysis of variance Alanine aminotransferase ALT AP Alkaline phosphatase aPTT Activated partial thromboplastin time Aspartate aminotransferase **AST AUC** Area under concentration-time curve Area under the plasma concentration-time curve from time zero to 24h  $AUC_{(0-24)}$ AUC<sub>(0-24)/D</sub> Dose-normalised AUC from time zero to 24h Area under the concentration-time curve from time zero to 24h  $AUC_{(0-24),norm}$ corrected by dose and body weight  $AUC_t$ AUC from time zero to time t  $AUC_{t-\infty}$ AUC from time t to infinity AUC from time zero (pre-dose) to the time of last quantifiable AUC<sub>t. norm</sub> concentration corrected by dose and body weight  $AUC_{\infty}$ Area under the plasma drug concentration vs. time from zero to infinity  $AUC_{\infty}/D$ The area under the plasma drug concentration vs. time curve from time zero to infinity, corrected for dose. The area under the concentration-time curve from time zero to infinity  $AUC_{\infty}$ , norm corrected by dose and body weight **BMI Body Mass Index** BP Blood pressure Below the limit of quantification **BQL** Confidence Interval CI CK Creatine kinase CL/F Apparent Total body clearance Maximum Plasma Concentration  $C_{max}$  $C_{max}/D$ C<sub>max</sub> corrected by dose C<sub>max</sub> corrected by dose and body weight  $C_{max,norm}$ Case Report Form **CRF** CTR Clinical Trial Report Coefficient of Variation CVBetween subject CV CVb ECG Electrocardiogram Glutamate dehydrogenase **GLDH** GGT Gamma-glutamyl transpeptidase HbA1C Glycated haemoglobin High-density lipoprotein **HDL** Hammersmith Medicines Research **HMR** HR Heart Rate International Conference on Harmonization **ICH** Investigational Medicinal Product **IMP** Immediate release IR Lactate dehydrogemnase LDH Low-density lipoprotein LDL Liquid Service Formulation LSF

**MCH** Hemoglobin amount per red blood cell The amount of hemoglobin relative to the size of the cell (hemoglobin **MCHC** concentration) per red blood cell **MCV** Average red blood cell size Medical Dictionary for Regulatory Activities MedDRA **MRT** Mean residence time Number of subjects N Number of observations used in analysis n PC Personal Computer Potential clinical importance **PCI** Pharmacodynamic(s) PD PK Pharmacokinetic(s) Portion of the ECG from the beginning of the P wave to the beginning PR of the QRS complex, representing atrioventricular node function. PT Prothrombin time O1 Lower quartile Q3 Upper quartile The QRS complex of the ECG reflects the rapid depolarization of the ORS right and left ventricles. QT Portion of the ECG between the onset of the Q wave and the end of the T wave, representing the total time for ventricular depolarization and repolarization. Corrected portion of the ECG between the onset of the Q wave and the QTc end of the T wave, representing the total time for ventricular depolarization and repolarization. OTc interval with Bazett's correction method **OTcB QTcF** QTc interval with Fridericia's correction method **RBC** Red blood cells RR Portion of the ECG between consecutive R waves, representing the ventricular rate SAP Statistical Analysis Plan SD Standard deviation Terminal elimination half-life  $t_{1/2}$ Dominant half-life  $t_{1/2,dom}$ **TEAE** Treatment-Emergent Adverse Event Time to maximum plasma concentration  $T_{max}$ Thyroid-stimulating hormone TSH Vz/FApparent volume of distribution WBC White blood cells

WHO

World Health Organisation

### 3 Introduction

This Statistical Analysis Plan (SAP) is based on the current trial protocol (version 5, Final 18 January 2017). Where statistical methods differ substantially between this SAP and the protocol, the differences will be identified in the SAP.

This SAP describes the datasets and the statistical methods to be used for the reporting and analysis of all data collected in Part 2 (cohorts 9 and 10), except for the 12-lead ECG continuous monitoring data which will be analysed by iCardiac Ltd (or an alternative provider), if applicable.

The randomisation code will not be broken before this SAP is finalised and signed. If a future protocol amendment necessitates a substantial change to the statistical analysis of the trial data, this SAP will be amended accordingly. If, after database lock, additional analyses are required to supplement the planned analyses described in this SAP, those unplanned analyses will not be described in an amended SAP, but they will be identified in the integrated clinical trial report (CTR). Any deviations from this SAP will be documented in the CTR.

This SAP has been written in consideration of the following guidelines:

- International Conference on Harmonization (ICH) E9, Guidance for Industry: Statistical Principles for Clinical Trials (ICH E9 1998)<sup>1</sup>; and
- ICH E3, Guidance for Industry: Structure and Content of Clinical Study Reports (ICH E3 1995)<sup>2</sup>.

Pharmacokinetic analysis will be done using WinNonlin v6.3 on a Windows PC. Statistical analysis will be done using SAS® 9.3 on a Windows PC.

# 4 Study Objective(s) and Endpoint(s)

### 4.1 Study Objective(s)

#### 4.1.1 Primary Objective(s)

• To investigate the safety and tolerability of emodepside (BAY 44-4400) after single oral doses administered as solution or immediate release (IR) tablets in healthy male subjects.

### 4.1.2 Secondary Objective(s)

• To investigate the pharmacokinetics (PK) of emodepside (BAY 44-4400), after administration as oral solution, and IR tablet (optional)

- To conduct an exploratory investigation of the relative bioavailability of the 5 mg and 20 mg IR tablet formulation using data generated in this study (optional)
- Possibility to determine the effect of food on the bioavailability of emodepside (BAY 44-4400) after single oral doses administered as solution or IR tablets.

## 4.2 Study Endpoint(s)

### 4.2.1 Safety and Tolerability Variables:

- Adverse Events (AEs).
- Physical and Neurological examination findings (including assessments of alertness, speech, language, and comprehension; cranial nerves; motor exam; coordination/cerebellar function; tremor of the hands, legs and head (postural, kinetic and rest tremor); sensation; and gait and postural stability (Pull test); mood; and sleepiness.).
- Vital signs: heart rate (HR), systolic and diastolic blood pressure (BP) in supine and sitting position (Cohort 10 only in supine), weight, body mass index (BMI; height at screening only), oral temperature.
- 12-lead ECG (HR, PR, QRS, QTcF), and for selected cohorts 12-lead ECG continuous recording (for emodepside exposure response analysis HR, PR, QRS and QTcF).
- Clinical laboratory parameters:
   <u>Hematology</u>: hemoglobin, hematocrit, MCV, MCH, MCHC, platelets, reticulocytes, white blood cells (WBC) differential, red blood cells (RBC), glycated haemoglobin (HbA1C) (at screening);
  - Coagulation: activated partial thromboplastin time (aPTT), prothrombin time (PT);
- <u>Biochemistry</u>: aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP), glutamate dehydrogenase (GLDH), gamma-glutamyl transpeptidase (GGT), LDH, CK, amylase, lipase, free T4 and T3, thyroid-stimulating hormone (TSH), glucose, cholesterol (high-density lipoprotein [HDL], and low-density lipoprotein [LDL], total), triglycerides, creatinine, urea, uric acid, bilirubin (total and conjugated), total protein, sodium, potassium, calcium, chloride and magnesium in serum;

• <u>Urinalysis</u>: by dipstick - glucose, ketone bodies, specific gravity, occult blood, pH, proteins, leucocytes, bilirubin, urobilinogen, nitrites.

• Ophthalmological assessments (Cohort 10 only)

#### 4.2.2 Pharmacokinetic Variables:

Based on the plasma concentration time data, the following PK parameters of emodepside will be calculated.

- Main PK parameters: AUC<sub>∞</sub>, AUC<sub>∞</sub>/D, C<sub>max</sub>, C<sub>max</sub>/D, of emodepside (BAY 44-4400)
- Exploratory PK parameters:  $C_{max,norm}$ ,  $T_{max}$ ,  $t_{1/2}$ , MRT, CL/F,  $AUC_{\infty,norm}$ ,  $AUC_{t}$ ,  $AUC_{t,norm}$ ,  $V_{z}/F$  of emodepside (BAY 44-4400)
- Other parameters:  $\lambda_z$ , AUC<sub>t- $\infty$ </sub>, points terminal

The following PK parameters of metabolites of emodepside may be calculated:  $AUC_{\infty}$ ,  $AUC_{\infty}/D$ ,  $C_{max}$ ,  $C_{max}/D$ ,  $C_{max,norm}$ ,  $T_{max}$ ,  $T_{1/2}$ ,  $AUC_{\infty,norm}$ ,  $AUC_{t}$ ,  $AUC_{t,norm}$ 

In urine, the amount and concentration of emodepside and possibly its metabolites will be measured. The appropriate specific PK parameters to be calculated will be decided according to the concentration.

#### 4.2.3 Pharmacodynamic Variables:

- Profiles of glucose and insulin, glucagon and cortisol (Cohort 9 only), only on Pre-Day (Day -1), Profile Day (Day 0), and Day 1.
- Single samples of prolactin and leptin, only on Pre-Day (Day -1), Profile Day (Day 0), and Day 1(Cohort 9 only).

# 4.3 Statistical Hypotheses

No formal statistical testing will be done.

# 5 Study Design

This is a single-center, blinded, randomised, placebo-controlled, parallel-group, single-dose, 2-cohort, dose-escalation, comparison study investigating safety, tolerability, and PK of

emodepside, after administration as an oral liquid service formulation (LSF) solution in healthy male subjects. Within each cohort, subjects will be randomised to receive either emodepside or placebo (n=8 per cohort; 6 assigned to emodepside and 2 assigned to placebo).

Subjects in Cohort 9 will receive 10mg solution of emodepside or matching placebo in a fed state and subjects in Cohort 10 will receive 40mg solution of emodepside in fasted state.



Table 1: Time and Events Table (Part 2, Cohort 9)

| Study Procedure | Screen | | | | | | | | | | | | | | | In-P | atien | t Pha | asea | | | | | | | | | | | | | | | T | ıble <sup>b</sup> | Follow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | | | | | | Pre | -Day | | | | | | | | | | Pro | file-l | Day | | | | | | | | Eva | luat | ion | | | 3 | ee 1a | bie " | Up |
| Day<br>± allowable deviation | -28 to -2 | -2 | | | | | • | -1 | | | | | | | | | | | 0 | | | | | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | | | | 7<br>+3 |
| Subject information and Informed Consent | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Medical history (including demographics and previous / concomitant medications) | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical examination <sup>c</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | Χ |
| Neurological examination <sup>d</sup> | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | Χ |
| Ward Admission (approx.16h) | | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Urine drugs of abuse and alcohol breath test | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Hours <sup>a</sup> (pre/post drug) | | -36 | -24° | -23.5 | -23 | -22. | -22 | -21 | -20 | -18 | -16 | -12 | 0* | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 5 | 6 | 8 | 12 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | | | | |
| Glucose, Insulin, Glucagon, and Cortisol profiles | | | Х | | Х | | Х | | Χ | | | X | Χ | | X | | Х | | | Х | | | | Х | Χ | | | | | | | | | | | |
| Samples for Prolactin & Leptin | | | Х | | | | | | | | | | X | | | | | | | | | | | | Χ | | | | | | | | | | | |
| Administration of emodepside <sup>e</sup> | | | | | | | | | | | | | Х | | | | | | | | | | | | | | | | | | | | | | | |
| 12-lead safety ECG <sup>f</sup> | Х | | Xf | Х | Χ | Х | Χ | Χ | Χ | | Χ | X | Χ <sup>f</sup> | X | Χ | Χ | Χ | | Χ | Χ | | | Χ | Χ | Χ | | Χ | Χ | Χ | Χ | Χ | Х | | | | Х |
| ECGs extracted from continuous recordings <sup>9</sup> | | | | | | | | | | | | | Xg | Xg | Xg | Xg | Χg | Χg | Xg | Χg | | Χ <sup>g</sup> | Xg | Χg | Χg | | | | | | | | | | | |
| Vital signs <sup>h</sup> | Х | | X <sup>h</sup> | Χ | Х | Х | X <sup>h</sup> | Χ | Xh | Х | Χ | X <sup>h</sup> | X <sup>h</sup> | Х | Χ | Χ | X <sup>h</sup> | | Χ | $X^h$ | | Χ | Χ | X <sup>h</sup> | $\chi^h$ | Х | Χ | Χ | Χ | Χ | Χ | Х | | | | Х |
| Adverse event monitoring | Χ | Χ | Χ | | | | Χ | | Χ | | | Χ | Χ | | Χ | | Χ | | Χ | Χ | | Χ | Х | Х | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | | | | Х |
| PK and metabolites <sup>j</sup> in plasma | | | | | | | | | | | | | χ <sup>j</sup> | Х | X <sup>j</sup> | Χ | $X^{j}$ | Χ | Χ | X <sup>j</sup> | | Х | X <sup>j</sup> | X <sup>j</sup> | $X^{j}$ | Χ | $X^{j}$ | Х | Х | Х | Χ | Χ | | | | Х |
| PK in urine <sup>k</sup> | | | | | | | | | | | | | | l | | 0–4 <sup>k</sup> | | | | | 4–8 <sup>k</sup> | | 8–12 <sup>k</sup> | 12–24 <sup>k</sup> | | | | | | | | | | | + | + |
| Laboratory Safety <sup>l,m</sup> | X m | | Х | | | 1 | | | | | | | Х | | | ٠, | | | | | Τ, σ | | 7 12 | | Х | | Х | Х | Χ | Х | Χ | Х | | | + | Х |
| Neurological <sup>d</sup> examination and short physical examination <sup>c</sup> | | | X° | | | | Х | | Х | | | Х | Х | | | | х | | | Х | | | | Х | Х | Х | Х | , , | | | | | | | | |

<sup>\*:</sup> In fasted subjects, all assessments at Hour –24 on Day –1 and Hour 0 on Day 0 are immediately before the administration of study drug (emodepside). In fed subjects, all assessments at Hour –24 on Day –1 and at Hour 0 on Day 0 are before the FDA breakfast. The only exception is the 12-lead ECG continuous recording (see footnote g).

<sup>&</sup>lt;sup>a</sup>: Including a 10-minute supine phase before supine BP, HR, body temperature, ECG; and for 5 minutes after each nominal timepoint for ECGs extracted from continuous recording (see footnote); and also recommended before drawing blood samples. Before sitting BP assessments minimum 3-minute sitting period.

b: If mean half-life of emodepside in any cohort is longer than predicted, there are options to extend in-house period, or out-patient ambulatory visits up to Day 14 if necessary, from Cohort 5 onwards and in subsequent cohorts. Refer to Option 1, Option 2, and Option 3 as outlined in Table .

Sponsor code: DNDI-EMO-001 Part 2

- c: Height at screening only, for calculation of BMI. Weight at screening for calculation of BMI, also at -24h (Day -1) for PK calculations.
- d: Neurological examination designed for the study, see Protocol Section 8.19.4 and Study Procedures Manual
- e: Administration of study drug while fasting or after a high-calorie, high-fat breakfast
- f: To include 3 repeat ECGs at these timepoints, with a time difference of about 1 minute, and single recordings at other timepoints
- <sup>9</sup>: For selected cohorts in Part 1 (see Protocol Section 8.19.2 continuous 12-lead ECG recording will be started 1 hour before dosing and continue for 24 hours post-dosing. ECGs will be extracted at predose, at three timepoints (-60, -45, and -30 minutes for fasted subjects or -90, -75, and -60 minutes for fed subjects) and at the timepoints at which PK blood samples are drawn. Subjects will be supine for 10 minutes prior to and 5 minutes after each nominal timepoint. When ECG extraction coincide with safety ECGs, vital signs and blood draws, procedures will be performed in said order.
- h: Vital signs to include BP (supine; plus sitting BP at the indicated timepoints<sup>th</sup>) and HR. Oral temperature only at screening and -24h.
- Exercise 4. Adverse Event (AE) monitoring will be throughout the study (spontaneous and solicited) to include questioning for tolerability and safety, however at these indicated timepoints will be specific questioning about AEs.
- In addition to the PK sample, metabolite samples are collected only for the indicated time points <sup>1</sup>. As an option, at the sponsor's discretion, an additional sample of no more than 1mL may be taken at each PK timepoint from all subjects in up to 2 cohorts.
- k: Start and end of urine collection for each bottle are indicated as hours post drug...
- Hematology, Coagulation, Chemistry: Urinalysis by dip stick.
- ": At Screening only: HIV 1, 2, Hepatitis B, C, HbA1C, in additional to hematology, coagulation, urinalysis, and chemistry.

Table 2. Follow-Up after Day 7 – Schedule Options 1, 2, or 3 Depending on Emodepside Plasma Concentrations at Day 7 in Previous Cohort(s) (from Cohort 5 onwards), Respectively.

For Screening and Days -2 through Day 8 see Table 1

| Г | T | | | | | |
|---|---|---|---|---|---|---|
| OPTION 1 | | | | Out-Patient Phase | | |
| Day | | | | | | Follow-Up Visit |
| | Discharge on Day 7 | | • | | | at 3 weeks (+3 days) post-dose |
| Physical Examination | , , | | | | | (see Table 1) |
| Neurological Examination | | | | | | (see Table 1) |
| 12-lead ECG | | | | | | (see Table 1) |
| Vital signs <sup>h</sup> | | | | | | (see Table 1) |
| Adverse event monitoring | | | | | | (see Table 1) |
| PK in plasma | | | | | | (see Table 1) |
| Laboratory Safety <sup>l,m</sup> | | | | | | (see Table 1) |
| OPTION 2 | | | | <b>Out-Patient Phase</b> | | |
| Day | Un to A via | to duni | ing the national from Day 9, 21 in | slucive (se needed) | | Follow-Up Visit |
| Day | - | | ing the period from Day 8–21 inc | ciusive (as needed) | | at 3 weeks (+3 days) post-dose |
| DI I I D | Ambulatory Evaluation Visits, S | chedul | ed As Needed | | | |
| Physical Examination | | | | | | (see Table 1) |
| Neurological Examination | | | | | | (see Table 1) |
| 12-lead ECG | | | | | | (see Table 1) |
| Vital signs <sup>h</sup> | | | | | | (see Table 1) |
| Adverse event monitoring <sup>1</sup> | X | | X | X | X | (see Table 1) |
| PK in plasma | X | | X | Χ | X | (see Table 1) |
| Laboratory Safety <sup>l,m</sup> | X | | X | Χ | X | (see Table 1) |
| OPTION 3 | | | Discharge from Ward on Day | X | | |
| _ | 8 (±1) | | 10 (±1) | 12 (±2) | 14 (±2) | |
| Day | (as needed) | | (as needed) | (as needed) | (max.) | Follow-Up Visit |
| | Prolonged In-House Evaluation | Phase | | / | | at 3 weeks (+3 days) post-dose |
| | with Discharge from Ward on D | | | | | ar o mono (15 aayo) poor acco |
| Physical Examination | | | | | | (see Table 1) |
| Neurological Examination | | | | | | (see Table 1) |
| 12-lead ECG | | | | | | (see Table 1) |
| Vital signs <sup>h</sup> | | | | | | (see Table 1) |
| Adverse event monitoring | X | | X | X | X | (see Table 1) |
| PK in plasma | X | | X | Χ | X | (see Table 1) |
| Laboratory Safety <sup>l,m</sup> | X | | X | Χ | X | (see Table 1) |

Table 3. Schedule of Events (Part 2, Cohort 10)

| Study Procedure | | ening<br>sits | | | | | | | | | | | | In-Patient Phase <sup>a</sup> | | | | | | | | | | | | | | | | t-pati | | it Follo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 1 | 2 | | | | | | Pre | -Da | у | | | | | | | | | Pro | ofile- | Day | | | | | | | I | Eva | luat | ion | | | ı | ohase | ' | w-Up |
| Day ± allowable deviation | -28 to<br>-2 | -7 to<br>-1 | -2 | | | | | | -1 | | | | | | 0 | | | | | | | | | | | 2 | 3 | 4 | 5 | 6 | 7 | 10<br>±1 | 14<br>±2 | 18<br>±2 | 21<br>+3 | | |
| Subject information and Informed Consent | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Medical history<br>(including<br>demographics,<br>previous/concomitant<br>medications) | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical examination <sup>b</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | Χ |
| Neurological examination <sup>c</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | Х |
| Colour blindness test <sup>d</sup> | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Ophthalmology exam <sup>e</sup> | | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | ı |
| Ward Admission (approx.16h) | | | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Urine drugs of abuse and alcohol breath test | Х | | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Hours <sup>a</sup> (pre/post<br>drug) | | | -36 | -24* | -23.5 | -23 | -22.5 | -22 | -21 | -20 | -18 | -16 | -12 | 0* | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 5 | 6 | 8 | 12 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | | | | |
| Glucose and Insulin profiles | | | | Х | | Х | | | | | | | X | X | | Χ | | | | | | | | | Х | Х | | | | | | | | | | | |
| Administration of emodepside <sup>f</sup> | | | | | | | | | | | | | | Х | | | | | | | | | | | | | | | | | | | | | | | |
| 12-lead safety ECG | Χ | | | Χ <sup>g</sup> | | Χ | | | | | | | X | Xg | | Χ | | | | | | | | | Χ | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | | | | Χ |
| Vital signs <sup>h</sup> | Χ | | | Χ | Χ | Χ | | | | | | X | Χ | Х | Χ | Χ | | | | | | | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | | | Χ |
| Adverse event monitoring <sup>i</sup> | Х | | Х | Х | | | | X | | X | | | X | Х | | Х | | Χ | | X | Χ | | Х | Х | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | Χ | Х |
| PK in plasma <sup>j</sup> | | | | | | | | | | | | | | Х | Χ | Χ | | | | (X) | | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ |
| Laboratory Safety <sup>k,l</sup> | Χ <sup>I</sup> | | | Χ | | | | | 1 | | | | | Х | | | | | | | | | | | | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Х | Х |
| Neurological <sup>c</sup> examination and short physical examination <sup>b</sup> | | | | X <sub>p</sub> | | Х | | | | | | | Х | Х | | Х | | | | | | | | | Х | Х | х | Х | | | | | | | | | |
| Travel and stay at ophthalmology clinic | | | | | | | | | | | | | | | | | Х | Χ | Χ | Х | Χ | Х | | | | | | | | | | | | | | | |
| Ophthalmology exam <sup>m</sup> | | | | | | | | | | | | | | | | | | | Χ | | | | | | | | | | | | | | | | <u> </u> | | |

<sup>\*</sup> All assessments at Hour 0 on Day 0 are immediately before the administration of study drug (emodepside), and assessments at Hour –24 on Day –1 will be time-matched to Profile Day

HMR code: 15-020 Part 2

Sponsor code: DNDI-EMO-001 Part 2

(dosing Day)

a Including a 10-minute supine phase before supine BP, HR, body temperature, ECG; and also recommended before drawing blood samples.

b Height at screening only, for calculation of BMI. Weight at screening for calculation of BMI, also at -24h (Day -1) for PK calculations.

<sup>&</sup>lt;sup>c</sup> Neurological examination designed for the study, see Protocol Section 8.19.4 and Study Procedures Manual.

<sup>&</sup>lt;sup>d</sup> Colour blindness to be determined at Screening visit 1.

e If subjects are eligible for study entry based on Screening visit 1 assessments, they will be asked to undergo an ophthalmology exam (Screening visit 2) within a week before Profile Day or on Pre—Day at the latest. All assessments for Screening Visit 1 will be performed prior to Screening Visit 2, but visits can be combined if necessary.

f Administration of study drug is in the fasted-state only.

<sup>&</sup>lt;sup>9</sup> To include 3 repeat ECGs at these timepoints, with a time difference of about 1 minute, and single recordings at other timepoints.

<sup>&</sup>lt;sup>h</sup> Vital signs to include supine BP and HR. Oral temperature only at screening and -24h.

Adverse Event (AE) monitoring will be throughout the study (spontaneous and solicited) to include questioning for tolerability and safety, however at these indicated timepoints will be specific questioning about AEs.

<sup>&</sup>lt;sup>j</sup> Timepoint shown as (X) indicates sample will be taken off-site whilst at the ophthalmology clinic. As an option, at the sponsor's discretion, an additional sample of no more than 1 mL may be taken at each PK timepoint from all subjects in up to 3 cohorts.

<sup>&</sup>lt;sup>k</sup> Hematology, Coagulation, Chemistry; Urinalysis by dip stick.

At Screening only: HIV 1, 2, Hepatitis B, C, HbA1C, in additional to hematology, coagulation, urinalysis, and chemistry.

<sup>&</sup>lt;sup>m</sup> Ophthalmology exams will be performed on Profile-Day (Day 0) approximately 2-2.5 h post-dose. If deemed necessary by the ophthalmologist additional ophthalmology follow-up visit(s) may be scheduled for eve-related AEs.

# 6 Planned Analyses

## 6.1 Interim Analyses

No interim analyses are planned. However, the blinded safety and PK data will be reviewed after Cohort 9.

#### **6.1.1** Persons responsible for analysis

Toni Mitchell (HMR) Statistician

Nick Jackson (HMR) SAS Programmer

## 6.2 Final Analysis

The database will be locked once all subjects have completed the study, data have been entered and all queries resolved. The final analysis will be carried out following database lock and unblinding.

#### 6.2.1 Persons responsible for analysis

Stephen Sah (HMR) Statistician

Nick Jackson (HMR) SAS Programmer

Bhavini Ladwa (HMR) Data Manager

# 7 Sample Size Considerations

# 7.1 Sample Size Assumptions

No formal sample size calculations have been performed as this is an exploratory study. A sample size of 8 per cohort will be considered sufficient to examine the safety and tolerability of emodepside as well as the PK after single oral administration of the investigational drug. For evaluation, a minimum number of 6 evaluable subjects per cohort is required.

HMR code: 15-020 Part 2

Sponsor code: DNDI-EMO-001 Part 2

# 8 Analysis Populations

The following population sets will be identified:

Safety Population: All subjects who received at least one dose of IMP.

PK Concentration Population: All subjects who received at least one dose of IMP and for

whom a pharmacokinetic sample has been analysed.

PK Parameter Population: All subjects in the PK Concentration Population for whom

pharmacokinetic parameters can be derived.

In all populations, treatment will be assigned based upon the treatment subjects actually received, regardless of the treatment to which they were randomised.

The primary endpoint will be analysed using the safety population.

### 8.1 Analysis Datasets

All analysis datasets will be based on observed data, except as outlined in Section 10.2.

# 9 Treatment Comparisons

The treatment comparison of interest is active (emodepside) versus placebo.

# 9.1 Data Display Treatment and Other Subgroup Descriptors

The sort order for treatment groups will be placebo, then study treatment in ascending dose order.

Listings of data will be sorted and displayed by treatment group, subject number, and also by date and time if applicable.

All subjects in cohorts 9 and 10 receiving the same formulation of placebo will be combined to form a pooled placebo group.

The treatment descriptions to be used on all tables and listings are:

Treatment GroupsShort DescriptionPlacebo [solution](Fed)PLA [sol](Fed)Placebo [solution](Fasted)PLA [sol](Fasted)Emodepside (xx mg) [solution](Fed)xx mg [sol](Fed)Emodepside (xx mg) [solution](Fasted)xx mg [sol](Fasting)

#### 9.1.1 Conventions for Summary Statistics and Data Displays

The minimum set of summary statistics for numeric variables will be: n, mean, standard deviation (or standard error), median, minimum, and maximum. 95% confidence intervals will be presented where appropriate for data interpretation.

Categorical data will be summarised in frequency tables with n and percentage. Summaries of a categorical variable will include all recorded values.

The minimum and maximum values will be presented with the same number of decimal places as the raw data collected on the CRF (or to 3 significant figures for derived parameters). The mean and percentiles (e.g. median, Q1, and Q3) will be presented using one additional decimal place. The standard deviation and standard error will be presented using two additional decimal places.

Placebo subjects will be pooled across cohorts 9 and 10 taking into account formulation and fed/fasted status.

# 10 Data Handling Conventions

### 10.1 Premature Withdrawal and Missing Data

All subjects who withdraw prematurely from the study or study drug will be included in the statistical analyses.

If a subject completes the treatment period but has missing data, then this will be made apparent in the subject listings. Missing data will not be imputed except for as outlined in Section 10.2.

If the study is prematurely discontinued, all available data will be listed and a review will be carried out to assess which statistical analyses are still considered appropriate.

Data collected at unscheduled time points during the study will not be used in the summaries or data analyses. They will be included in the listings.

If time information (i.e. hours and/or minutes) for adverse events or concomitant medication is missing, but the day is present, then the time will be calculated in days. If date information is partial or missing, then any derived times (e.g. AE start time from last study medication) will be listed as missing.

Conventions for handling missing plasma concentrations are given in Appendix B.

#### 10.2 Derived and Transformed Data

For ECGs, vital signs, glucose, insulin, glucagon, cortisol and neurological examinations recorded on Day -1 the baseline will be the -24 h value and for Day 0 the baseline will be the pre-dose value on Day 0. The AUC<sub>0-24</sub> for change from baseline in glucose, insulin, glucagon and cortisol will be calculated on Day -1 and Day 0, using the linear-linear trapezoidal method. For prolactin and leptin the baseline will be pre-dose on Day 0.

Laboratory data will be reported in standard units. The baseline will be the latest value recorded pre-dosing on Day 0. Out-of-range laboratory tests may be repeated. If a test is out-of-range at a baseline timepoint and repeated before dosing, the latest repeat value before dosing will be used as baseline. However, if a test is out-of-range and repeated at any other time during the study, the out-of-range value (not the repeat value) will be included in statistical summaries.

Triplicate ECG measurements will be made at some timepoints on Day -1 and Day 0, the mean of the three measurements for each subject will be used at each timepoint.

The pharmacokinetic parameters to be derived are given in Appendix B

#### 10.3 Assessment Windows

No assessment windows are defined for this report.

### 10.4 Values of Potential Clinical Importance

Any laboratory value outside the reference interval for that variable will be flagged with an 'H' if it is higher than the reference interval, and with an 'L' if it is lower. Additionally, if, during the course of the trial, a variable changes from baseline (Day 0) by more than a predetermined amount (as defined by the Principal Investigator, Appendix A), that value will receive a flag 'I' if increased, or 'D' if decreased. Therefore, if a value both falls outside the reference interval and alters from the baseline value by more than the predetermined amount, it will attract a double flag and will be considered to be potentially clinically important.

A vital signs result will be considered to be of potential clinical importance if it falls outside the relevant range below:

| Vital Sign | Range |
|------------------------------------------------|------------------|
| Supine/semi-recumbent systolic blood pressure | 85–160 mm Hg |
| Supine/semi-recumbent diastolic blood pressure | 40–90 mm Hg |
| Supine/semi-recumbent heart rate | 40–100 beats/min |
| Respiration rate | 8–20 per min |
| Oral temperature | 35.5–37.8°C |

QTcB or QTcF > 450 msec and increases in QTcB or QTcF from baseline of > 30 msec will be considered to be potentially clinically important.

# 11 Study Population

### 11.1 Disposition of Subjects

The disposition of all subjects in the safety population will be summarised including: number of subjects randomised; number completing the study (i.e. not withdrawn), by treatment; and number discontinued (withdrawn) from the study. The number of subjects in each analysis population will be summarised by treatment.

All subjects who withdraw or are withdrawn from the study will be listed, by treatment, with the reason for withdrawal.

A listing of analysis populations will be provided.

#### 11.2 Protocol Deviations

Before closing the database, data listings will be reviewed to identify any significant deviations and determine whether the data should be excluded from any analysis populations.

Major protocol deviations include subjects who:

- Entered the study even though they did not satisfy the entry criteria.
- Met the criteria for withdrawal from the study but were not withdrawn.
- Received the wrong treatment or incorrect dose.
- Received an excluded concomitant therapy.
- Received investigational product(s) past the expiration date and time.

• Had their treatment assignment unblinded.

In addition, subjects with minor time deviations (measurements taken outside the allowable windows given in the protocol) will be identified.

### 11.3 Demographic and Baseline Characteristics

Demographic and baseline characteristics (e.g. physical examination, neurological examination, vital signs and ECGs) will be listed and summarised.

Subjects who take concomitant medication will be listed. All non-trial medication will be coded using version September 2016 of the WHO Drug dictionary.

### 11.4 Treatment Compliance

Dates and times of dosing will be listed.

# 12 Safety Analyses

Summaries and listings of safety data will use the safety population.

## 12.1 Extent of Exposure

The dates and times of treatment dosing will be listed to indicate exposure to the study medication.

#### 12.2 Adverse Events

Adverse events will be coded using the version of the Medical Dictionary for Regulatory Activities (MedDRA) (version 20.0).

All adverse events will be listed.

The number of subjects with at least one treatment-emergent adverse event (TEAE) will be tabulated by actual treatment and MedDRA system organ class and preferred term. A treatment-emergent adverse event is defined as an event emerging during treatment having been absent pre-treatment or having worsened relative to pre-treatment<sup>1</sup>.

For each of the following, the number of subjects with adverse events will be summarised by actual treatment:

TEAEs by system organ class and preferred term

• Drug-related ("related" as recorded by the Investigator) TEAEs by system organ class and preferred term

Subjects with more than one TEAE will be counted only once, at the greatest severity or causal relationship, for each system organ class and preferred term. Adverse events with missing severity and/or causality will be treated as severe and related, respectively.

Summaries will be sorted by system organ class and decreasing total incidence of preferred term.

#### 12.3 Deaths and Serious Adverse Events

Adverse events leading to deaths and serious adverse events will be listed separately (fatal events will be listed separately from non-fatal events).

### 12.4 Adverse Events Leading to Withdrawal from the Study

Adverse events leading to withdrawal will be listed separately.

### 12.5 Clinical Laboratory Evaluations

Haematology, clinical chemistry and urinalysis evaluation at each planned assessment, and change from baseline at each planned post-baseline assessment, will be summarised by actual treatment.

Urinalysis parameters will also be listed.

All laboratory values of potential clinical importance will be listed and all related laboratory results (i.e. haematology or clinical chemistry) for subjects with values of potential clinical importance will be listed, separately. Frequencies of laboratory values of potential clinical importance will be summarised.

### 12.6 Other Safety Measures

#### 12.6.1 Vital signs

Vital signs evaluation at each planned assessment, and change in vital signs baseline at each planned post-baseline assessment, will be summarised by actual treatment. Individual subject profiles will be plotted for each vital sign parameter (Blood Pressure and Heart Rate).

Vital signs data of potential clinical importance will be listed separately.

#### 12.6.2 ECG

QT interval data will be presented using Bazett's (QTcB) and Fridericia's (QTcF) corrections.

ECG data will be summarised by treatment and time point. Differences from baseline will be summarised by treatment and time point.

The number of subjects with a potentially clinically important ECG value will be summarised by actual treatment and time point, giving the numbers of subjects with QT, QTcB or QTcF > 450 msec, > 480 msec and > 500 msec, and the numbers of subjects with increases in QT, QTcB or QTcF from baseline of > 30 msec and > 60 msec<sup>3</sup>. A supporting listing of all subjects with an ECG value of potential clinical importance and a separate listing of ECG findings classified as abnormal by the Investigator will also be provided.

#### 12.6.3 Neurological examination

Neurological examination results will be summarised and normal and abnormal neurological examination findings will be listed in detail according to the CRF. Total scores from neurological questionnaires at each planned assessment, and change from baseline at each planned post-baseline assessment, will be summarised by actual treatment.

Total scores from neurological questionnaires will also be listed.

## 12.6.4 Physical examination

Physical examination results will be summarised and abnormal physical examination findings will be listed.

#### 12.6.5 Ophthalmology assessments

Ophthalmology assessments results will be summarised and listed by time point.

# 13 Pharmacokinetic Analyses

Analytical Services International Ltd, London, U.K. will measure the plasma and urine concentrations of emodepside. The pharmacokinetic analysis will be done by Statistics and Data Management Department at HMR. Pharmacokinetic parameters will be calculated using WinNonlin, version 6.3.

In addition, the plasma and urine concentration of emodepside metabolite(s) may be measured. If and when these data become available a SAP amendment will be written to specify their reporting (if applicable).

The pharmacokinetic parameters to be derived are given in Appendix B.

PK concentration data will be summarised using the PK concentration population. PK parameters will be summarised using the PK Parameter population.

For log transformed parameters, the primary measure of central tendency will be the geometric mean<sup>4</sup>; for untransformed parameters, it will be the arithmetic mean or median.

For all variables N (number of subjects receiving the treatment/formulation in the population), n (number of observations), arithmetic mean, median, minimum, maximum, SD, %CV, and the 95% confidence interval for the arithmetic mean will be provided. For log-transformed variables, all of the above plus the geometric mean, which is the anti-logged arithmetic mean of log-transformed variables, its 95% confidence interval and the SD of the logs will be provided.

The between-subject CV will be calculated using:

- 1. %CVb = 100 \* (SD/Mean) with SD and Mean of untransformed data
- 2. %CVb =  $100 * \sqrt{(\exp(SD)^2 1)}$  with SD of log-transformed data

### 13.1 Plasma PK

#### 13.1.1 Pharmacokinetic Concentration Data

The plasma concentrations of emodepside and metabolites (if applicable) will be listed and summarised by treatment. Means at any time will only be calculated if at least 2/3rds of the individual data points are above the lower limit of quantification.

Individual and mean plasma concentration—time profiles will be presented graphically.

#### 13.1.2 Pharmacokinetic Parameters

The pharmacokinetic parameters of emodepside and metabolites (if applicable) will be listed and summarised by treatment.

To assess the effect of food, analysis of variance (ANOVA) models will be fitted to the fed (Part 2, Cohort 9) solution and relevant fasted (Part 1, Cohort 5) solution data with the logarithm of the pharmacokinetic parameters  $AUC_{0-24}$  as the dependent variable, and formulation as a fixed effect. The estimated least square means and residual variance from the model will be used to construct 90% CIs for the difference in means on the log scale for the comparison of fed versus fasted solutions.

### 13.2 Urinary PK

If concentrations of emodespide in urine are determined, the amount of emodespide excreted in the urine will be estimated. The data will be listed and summarised by treatment.

# 14 Pharmacodynamic Analyses

Summaries and listings will use the safety population.

Pharmacodynamic variables (glucose, insulin, glucagon, cortisol, prolactin and leptin) at each planned assessment, and change from baseline at each planned post-baseline assessment, will be summarised by actual treatment.

In addition, for glucose and insulin (Cohorts 9 and 10), glucagon and cortisol (Cohort 9):

- Individual subject profiles will be plotted
- The difference between change from baseline on Day 0 and Day -1 will be summarised at each planned post-baseline assessment by actual treatment
- The AUC<sub>0-24</sub> of change from baseline will be summarised for each day and treatment

Individual Insulin and PK Concentration Plots, including Related Significantly Important AE Durations will be produced.

For calculation of pharmacodynamics parameters, summary statistics and individual profile plots, values below the quantifiable limit of the assay will be substituted by one half of the lower limit of quantification.

# 15 Changes from the Protocol Specified Statistical Analysis

After the study was submitted to the MHRA and ethics committee the following changes were made to the analyses:

- 1) The definition of treatment-emergent adverse event has been updated from "an AE will be considered as treatment emergent if it appeared after the first dosing, or if appeared before dosing and worsened after dosing" to:
  - A treatment-emergent adverse event is defined as an event emerging during treatment having been absent pre-treatment or having worsened relative to pre-treatment<sup>1</sup>.
- 2) The AUC<sub>0-24</sub> of change from baseline for glucose, insulin, glucagon and cortisol will be summarised for each day and treatment
- 3) The following emodepside parameters have been added to those mentioned in the protocol:

Main PK parameters: AUC<sub>0-24</sub> and AUC<sub>0-24</sub>/D

Exploratory PK parameters: AUC<sub>0-24</sub>,<sub>norm</sub> ,t<sub>1/2,dom</sub>

4) The following analyses have been added for glucose, insulin, glucagon and cortisol:

The difference between change from baseline on Day 0 and Day -1 will be summarised at each planned post-baseline assessment by actual treatment

The AUC<sub>0-24</sub> of change from baseline will be summarised for each day and treatment

#### 16 References

 International Conference on Harmonization, 1998. Statistical Principles for Clinical Trials - ICH Harmonised Tripartite Guideline. Guidance for Industry, E9, FDA federal register, Vol 63, 1998, p49583. Available at: http://www.fda.gov/cder/guidance.

2. International Conference on Harmonization, 1995. Structure and Content of Clinical Study Reports - ICH Harmonised Tripartite Guideline. Guidance for Industry, E3, FDA federal register, Vol 61, 1996, p37320. Available at: http://www.fda.gov/cder/guidance.

- International Conference on Harmonisation, 2005. Clinical Evaluation of QT/QTc
   Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs.
   Concept paper, Guidance for Industry, E14, Center for Drug Evaluation and Research (CDER). Available at: http://www.fda.gov/cder/guidance/6922fnl.htm.
- 4. Julious, SA & Debarnot, CAM (2000) "Why are Pharmacokinetic Data Summarised by Arithmetic Means?", Journal of Biopharmaceutical Statistics, 10 (1), p55-71.
- 5. FL140 HMR Laboratory alert and delta ranges ver 3 (HMR Lab form).

# 17 ATTACHMENTS

# 17.1 Table of Contents for Data Display Specifications

For overall page layout refer to Appendix C.

Tables, figures and listings will be labelled B for Part 2, e.g., 14.1B

The numbering in the tables below will take precedence over the numbering in the shells.



The following tables and figures will be produced (templates provided in Sections 17.2.1 and 17.2.2):

| Table | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 10.1 | Summary of Subject Disposition | Safety | 16.2.1.2, | T_SD1 |
| | | | 16.2.3.1 | |
| 14.1 | DEMOGRAPHIC DATA | | | |
| 14.1 | Summary of Demographic Characteristics | Safety | 16.2.4.1 | <u>T_DM1</u> |
| 14.2 | PHARMACOKINETIC AND PHARMACODYNAMIC | | | |
| | DATA | | | |
| 14.2.1.1 | Summary of Emodepside Plasma Pharmacokinetic | PK | 16.2.6.1.1 | <u>T_PK1</u> |
| | Concentration-Time Data (ng/mL) | | | |
| 14.2.1.2 | Summary of Derived Emodepside Plasma Pharmacokinetic | PK | 16.2.6.1.2 | <u>T_PK3</u> |
| | Parameters | | | |
| 14.2.1.3 | Summary of Log-Transformed Derived Emodepside Plasma | PK | 16.2.6.1.2 | <u>T_PK4</u> |
| | Pharmacokinetic Parameters | | | |
| 14.2.1.4 | Assessment of the Effect of Food on the PK of Emodepside | PK | 16.2.6.1.2 | <u>T_PK7</u> |
| 14.2.2 | Summary of Derived Emodepside Urine Pharmacokinetic | PK | 16.2.6.2 | <u>T PK3</u> |
| | Parameters | | | _ |
| 14.2.3.1 | Summary of Glucose | Safety | 16.2.6.3 | T_PD1 |
| 14.2.3.2 | Summary of Difference Between Day -1 and Day 0 in | Safety | 16.2.6.3 | <u>T_PD2</u> |
| | Glucose | | | |
| 14.2.3.3 | Summary of AUC <sub>0-24</sub> for Change from Baseline in Glucose | Safety | 16.2.6.4 | <u>T_PD3</u> |
| 14.2.4.1 | Summary of Insulin | Safety | 16.2.6.3 | <u>T_PD1</u> |
| 14.2.4.2 | Summary of Difference Between Day -1 and Day 0 in Insulin | Safety | 16.2.6.3 | T_PD2 |
| 14.2.4.3 | Summary of AUC <sub>0-24</sub> for Change from Baseline in Insulin | Safety | 16.2.6.3 | <u>T_PD3</u> |
| 14.2.5.1 | Summary of Glucagon | Safety | 16.2.6.3 | <u>T_PD1</u> |
| 14.2.5.2 | Summary of Difference Between Day -1 and Day 0 in | Safety | 16.2.6.3 | <u>T_PD2</u> |
| | Glucagon | | | |
| 14.2.5.3 | Summary of AUC <sub>0-24</sub> for Change from Baseline in Glucagon | Safety | 16.2.6.3 | T_PD3 |

| Table | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 14.2.6.1 | Summary of Cortisol | Safety | 16.2.6.3 | T_PD1 |
| 14.2.6.2 | Summary of Difference Between Day -1 and Day 0 in | Safety | 16.2.6.3 | <u>T_PD2</u> |
| | Cortisol | | | |
| 14.2.6.3 | Summary of AUC <sub>0-24</sub> for Change from Baseline in Cortisol | Safety | 16.2.6.3 | T_PD3 |
| 14.2.7 | Summary of Prolactin | Safety | 16.2.6.3 | <u>T_PD1</u> |
| 14.2.8 | Summary of Leptin | Safety | 16.2.6.3 | <u>T_PD1</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Summary of Treatment-Emergent Adverse Events | Safety | 16.2.7.1 | T AE1 |
| 14.3.1.2 | Summary of Drug-Related Treatment-Emergent Adverse Events | Safety | 16.2.7.1 | T_AE1 |
| 14.3.1.3 | Summary of Treatment-Emergent Adverse Events by Severity Grade | Safety | 16.2.7.1 | T_AE1 |
| 14.3.1.4 | Summary of Drug Related Treatment-Emergent Adverse<br>Events by Severity Grade | Safety | 16.2.7.1 | T_AE1 |
| 14.3.2.1 | Listing of Fatal Adverse Events | Safety | 16.2.7.1 | L AE1 PG |
| 14.3.2.2 | Listing of Non-Fatal Serious Adverse Events | Safety | 16.2.7.1 | L AE1 PG |
| 14.3.2.3 | Listing of Other Significant Adverse Events | Safety | 16.2.7.1 | L AE1 PG |
| 14.3.3 | Narratives of deaths, other serious and significant adverse events | Safety | | - |
| 14.3.4 | Summary of Laboratory Values of Potential Clinical Importance | Safety | 16.2.8.1,<br>16.2.8.3 | <u>T_LB1</u> |
| 14.3.5.1 | Summary of Chemistry Laboratory Values | Safety | 16.4 | T LB2 |
| 14.3.5.2 | Summary of Haematology Laboratory Values | Safety | 16.4 | <u>T_LB2</u> |
| 14.3.5.3 | Summary of Urinalysis Dipstick Results | Safety | 16.2.8.5 | T UR1 |
| 14.3.6.1 | Summary of Vital Signs | Safety | 16.4 | T_VS1 |
| 14.3.6.2 | Summary of AUC0-24 for Change from Baseline in Supine Diastolic Blood Pressure (h*mmHg) | Safety | 16.4 | <u>T_VS2</u> |
| 14.3.6.3 | Summary of AUC0-24 for Change from Baseline in Supine Systolic Blood Pressure (h*mmHg) | Safety | 16.4 | <u>T_VS2</u> |
| 14.3.6.4 | Summary of AUC0-24 for Change from Baseline in Supine | Safety | 16.4 | <u>T_VS2</u> |

| Table | Description | Population | Source<br>Listing | Template<br>(Shells below) |
|---|---|---|---|---|
| | Heart Rate (h*beats/min) | | | |
| 14.3.7.1 | Summary of ECG values | Safety | 16.4 | T_EG2 |
| 14.3.7.2 | Summary of ECG Values and Changes in ECG Values of | Safety | 16.4 | T_EG3 |
| | Potential Clinical Importance | | | |
| 14.3.8.1 | Summary of Neurological Examination Data | Safety | 16.2.9.5 | T_NE1 |
| 14.3.8.2 | Summary of Neurological Examination Questionnaire Data | Safety | 16.2.9.6 | T_LB2 |
| 14.3.9 | Summary of Physical Examination Data | Safety | 16.2.9.4 | <u>T_PE1</u> |
| 14.3.10 | Summary of Ophthalmological Examination Data | Safety | 16.2.9.7 | T NE1 |

| Figure | Description | Population | <b>Source Listing</b> | Template (Shells below) |
|---|---|---|---|---|
| 14.2 | PHARMACOKINETIC AND PHARMACODYNAMIC DATA | | | |
| 14.2.1.1 | Individual Emodepside Plasma Concentration-Time Plots (Linear and Semi-log) | PK | 16.2.6.1.1 | <u>F_PK1</u> |
| 14.2.1.2 | Geometric mean (+/- SD) Emodepside Plasma<br>Concentration-Time Plots (Linear and Semi-log) | PK | 16.2.6.1.1 | <u>F_PK2</u> |
| 14.2.2.1 | Individual Glucose-Time Plots | PD | 16.2.6.3 | <u>F_PD1</u> |
| 14.2.2.2 | Individual Glucose and PK Concentration Plots - | PD | 16.2.6.3, | |
| | Including Related Significantly Important AE Durations | | 16.2.6.1.1,<br>16.2.7.1 | F_PD2 |
| 14.2.3.1 | Individual Insulin-Time Plots | PD | 16.2.6.3 | <u>F_PD1</u> |
| 14.2.3.2 | Individual Insulin-Time Plots 0-12h | PD | 16.2.6.3 | F PD1 |
| 14.2.3.3 | Individual Insulin and PK Concentration Plots - | PD | 16.2.6.3, | F PD2 |
| | Including Related Significantly Important AE Durations | | 16.2.6.1.1, | |
| | | | 16.2.7.1 | |
| 14.2.4 | Individual Glucagon-Time Plots | PD | 16.2.6.3 | <u>F PD1</u> |
| 14.2.5 | Individual Cortisol-Time Plots | PD | 16.2.6.3 | <u>F_PD1</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Individual Systolic Blood Pressure-Time Plots | Safety | 16.2.9.1 | F_PD1 |
| 14.3.1.2 | Individual Diastolic Blood Pressure-Time Plots | Safety | 16.2.9.1 | F_PD1 |
| 14.3.2 | Individual Heart Rate-Time Plots | Safety | 16.2.9.1 | F PD1 |

The following abbreviated listings will be produced (templates provided in Section 17.2.3):

| Listing | Description | Template (Shells below) |
|---|---|---|
| 16.2.1 | Study dates & disposition of subjects | |
| 16.2.1.1 | Listing of Study Dates | L_SD1_PG |
| 16.2.1.2 | Listing of Reasons for Withdrawal | L SD2 PG |
| 16.2.2 | Protocol deviations | |
| 16.2.2.1 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | L DV1 PG |
| 16.2.2.2 | Listing of Subjects with Time Deviations | L_TD1_PG |
| 16.2.2.3 | Listing of Subjects with Other Protocol Deviations | L_DV2_PG |
| 16.2.3 | Analysis sets, including subjects excluded from analysis | |
| 16.2.3.1 | Listing of Analysis Populations | <u>L_AN1_PG</u> |
| 16.2.4 | Demographic data & concomitant medication | |
| 16.2.4.1 | Listing of Demographic Characteristics | L_DM1_PG |
| 16.2.4.2 | Listing of Concomitant Medications | L CM1 PG |
| 16.2.5 | Study drug administration | |
| 16.2.5.1 | Listing of Exposure Data | <u>L_EX1_PG</u> |
| 16.2.6 | Pharmacokinetic and Pharmacodynamic data | |
| 16.2.6.1.1 | Listing of Emodepside Plasma Pharmacokinetic Concentration-Time | L PK1 PG |
| | Data | <u>L_IKI_IU</u> |
| 16.2.6.1.2 | Listing of Derived Emodepside Plasma Pharmacokinetic Parameters | <u>L_PK4_PG</u> |
| 16.2.6.1.3 | Individual Emodepside Plasma Concentration-Time Plots (log scale) for | F PK10 |
| | Estimation of λz, with Regression Line | <del></del> |
| 16.2.6.2 | Listing of Emodepside Urine Excretion Rate Data | L PK3 PG |
| 16.2.6.3 | Listing of PD concentration-Time Data | L PK1 PG |
| 16.2.6.4 | Listing of Derived AUC0-24 PD Concentration-Time Data | <u>L_PK1_PG</u> |
| 16.2.7 | Adverse events | |
| 16.2.7.1 | Listing of All Adverse Events | L_AE1_PG |
| 16.2.7.2 | Listing of Serious Adverse Events | L_AE1_PG |

| 16.2.7.3 | Listing of Adverse Events Leading to Withdrawal from Study | L_AE1_PG |
|---|---|---|
| 16.2.8 | Laboratory values | |
| 16.2.8.1 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance | L_LB1_PG |
| 16.2.8.2 | Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities | L_LB2_PG |
| 16.2.8.3 | Listing of Haematology Abnormalities of Potential Clinical Importance | L LB1 PG |
| 16.2.8.4 | Listing of All Haematology Laboratory Data for Subjects with PCI Abnormalities | L_LB2_PG |
| 16.2.8.5 | Listing of Urinalysis Data | <u>L URI</u> |
| 16.2.9 | Vital signs, ECG variables, neurological, physical findings and Ophthalmological Assessment | |
| 16.2.9.1 | Listing of Vital Signs of Potential Clinical Importance | L VS1 PG |
| 16.2.9.2 | Listing of ECG Values of Potential Clinical Importance | L EG1 PG |
| 16.2.9.3 | Listing of Abnormal ECG Findings | L EG2 PG |
| 16.2.9.4 | Listing of Abnormal Physical Examination Findings | L PE1 PG |
| 16.2.9.5 | Listing of Neurological Examination Findings | L NE1 PG |
| 16.2.9.6 | Listing of Neurological Questionnaire Findings | L NE2 PG |
| 16.2.9.7 | Listing of Ophthalmological Examination Data | L NE1 PG |

Complete listings of all data collected in this study will also be produced.

HMR code: 15-020 Part 2

Sponsor code: DNDI-EMO-001 Part 2

# 17.2 Data Display Specifications

#### 17.2.1 Table Outlines

#### Template T\_SD1

Table 10.1 Summary of Subject Disposition

| Population | Status | Reason for Withdrawal | Treatment 1 | Treatment 2 | Etc | All Subjects |
|---|---|---|---|---|---|---|
| Safety Population | Randomised | | | | | |
| | Completed | | | | | |
| | Withdrawn | | | | | |
| | | Death | | | | |
| | | Adverse Events | | | | |
| | | Withdrawal by subject | | | | |
| | | Physician decision | | | | |
| | | Protocol violation | | | | |
| | | Study terminated by | | | | |
| | | Sponsor | | | | |
| | | Lost to follow-up | | | | |
| | | Other | | | | |
| PK Concentration | Included | | | | | |
| PK Parameter | Included | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and column for "All emodepside"

This table will contain one column for placebo, each dose/formulation, all active and all subjects.
### Template T\_DM1

Table 14.1 Summary of Demographic Characteristics

| Variable | Statistics | Treatment 1<br>(N=xx) | Treatment 2<br>(N=xx) | Etc | All Subjects (N=xx |
|---|---|---|---|---|---|
| Age (y) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |
| Sex | N | | | | |
| | Male | | | | |
| Race | American Indian or Alaskan | | | | |
| | Native | | | | |
| | Asian | | | | |
| | Black | | | | |
| | Native Hawaiian or other | | | | |
| | Pacific Islander | | | | |
| | White | | | | |
| | Other | | | | |
| Ethnicity | Hispanic or Latino | | | | |
| | Not Hispanic or Latino | | | | |
| Height (cm) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |
| Weight (kg) | n | | | | |
| | Mean | | | | |
| | SD | | | | |

| Variable | Statistics | Treatment 1<br>(N=xx) | Treatment 2<br>(N=xx) | Etc | All Subjects (N=xx) |
|---|---|---|---|---|---|
| | Min | (11 701) | (11 70) | | |
| | Median | | | | |
| | Max | | | | |
| BMI (kg/m2) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |
| Cigarettes* | n | | | | |
| (daily) | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |
| Alcohol* | n | | | | |
| (units/week) | Mean | | | | |
| | SD | | | | |
| | Min | | | | |
| | Median | | | | |
| | Max | | | | |

\*includes only those subjects who drink alcohol or smoke Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and additional demographic characteristics

#### Template T\_AE1

Table 14.3.3.xx Summary of Treatment-Emergent Adverse Events

| | | Treatme | nt 1 (N=xx) | Treatm | ent 2 (N=xx) | Etc |
|---|---|---|---|---|---|---|
| System Organ Class | Preferred Term | n | % | n | % | |
| Number of subjects with AEs | | | | | | |
| Gastrointestinal disorders | Total number of subjects | | | | | |
| | Abdominal discomfort | | | | | |
| | Abdominal pain | | | | | |
| | <b>↓</b> | | | | | |
| Nervous system disorders | Total number of subjects | | | | | |
| | Dizziness | | | | | |
| | Headache | | | | | |
| | <b>\</b> | | | | | |
| $\downarrow$ | $\downarrow$ | | | | | |

<sup>\*</sup>Subjects with ≥1 adverse event are counted only once per system organ class and preferred term.

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

SOCs and PTs are sorted in decreasing order of frequency

Presented for all applicable MedDRA system organ classes and terms. For tables by severity a sub-heading will be added to each table page

Sponsor code: DNDI-EMO-001 Part 2

#### Template T\_LB1

Table 14.3.4.xx Summary of Laboratory Values of Potential Clinical Importance

| | | Planned Relative | | Doub | le Flags |
|----------|--------------------|------------------|---|------|----------|
| Lab Test | Treatment | Time | n | HI | LD |
| | Treatment 1 (N=xx) | | | | |

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Source: Listing 16.2.xx

Programming notes: Continued with all tests, treatment groups and time points

#### Template T\_LB2

Table 14.3.3.2 Summary of Chemistry Laboratory Values

| | | | | | | | | | | | Cha | ange fr | om Baselin | ie | , |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned | | | | | | | | | | | | | |
| Laboratory Test (units) | Treatment | Relative Time | n | Mean | 95% CI | SD | Median I | Min | Max | n | Mean | SD | Median | Min | Max |
| | Treatment 1 (N=xx) | -20h | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all treatments and time points.

For the summary of neurological questionnaires the first column will be headed "Questionnaire (Total Score)" and the footnote will be removed

Sponsor code: DNDI-EMO-001 Part 2

#### Template T\_UR1

Table 14.3.3.4 Summary of Urinalysis Dipstick Results

| Planned Relative | | Treatm | ent 1 (N=xx) | Treatm | ent 2 (N=xx) |
|---|---|---|---|---|---|
| Flatilled Relative | | Treatin | CITC I (IV-XX) | ircatiii | CITE Z (IV-XX) |
| Time | Result | n | % | n | % |
| Time 1 | Positive | | | | |
| | Negative | | | | |
| | No Result | | | | |
| | Not Done | | | | |
| Time 2 | Positive | | | | |
| | Negative | | | | |
| | No Result | | | | |
| | Not Done | | | | |

Source: Listing 16.2.xx

Programming notes: Results recorded as received, e.g. Negative, Trace, etc; urine pH summarized as <5, 5-8, >8

Continued with all treatment groups and time points

#### Template T\_VS1

Table 14.3.4 Summary of Vital Signs

| | | | | | | | | | Chan | ge from Bas | eline | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned | | | | | | | | | | | | |
| | Treatment | Relative Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Systolic BP (mmHg) | Treatment 1 (N=xx) | -20h | | | | | | | | | | | | |

Source: Listing 16.2.xx

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all variables, treatments and time points.

### Template T\_VS2

Table 14.3.4 Summary of AUCO-24 for Change from Baseline in Supine Diastolic Blood Pressure (h\*mmHg)

| | | | Day | / -1 | | | | Day | 0 | | | | Day ( | 0 - Day -1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | Mean | SD | Min | Max | n | Mean | SD | Min | Max | N | Mean | SD | 95% CI (Lower, Upper) |
| Treatment 1 (N=xx) | | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Difference is change from mean baseline

Programming notes: Continued with all treatments

#### Template T\_EG2

Table 14.3.5.1 Summary of ECG Values

| | | | | | | | | | Char | ge from B | aseline | 9 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned Relative | | | | | | | | | | | | |
| Variable | Treatment | Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Heart Rate (bpm) | Treatment 1 (N=xx) | -20h | | | | | | | | | | | | |
| | | -21h | | | | | | | | | | | | |
| | | -23h | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | -20h | | | | | | | | | | | | |
| | | -21h | | | | | | | | | | | | |
| | | -23h | | | | | | | | | | | | |
| PR Interval (msec) | Treatment 1 (N=xx) | -20h | | | | | | | | | | | | |
| | | -21h | | | | | | | | | | | | |
| | | -23h | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | -20h | | | | | | | | | | | | |
| | | -21h | | | | | | | | | | | | |
| | | -23h | | | | | | | | | | | | |

Sponsor code: DNDI-EMO-001 Part 2

Source: Listing 16.2.xx

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all treatment groups and time points. Do not summarise RR or QRS axis

#### Template T\_EG3

Table 14.3.7.xx Summary of ECG Values and Changes in ECG Values of Potential Clinical Importance

| | | Planned<br>Relative | 451 – 48 | 30 msec | 481, – 500 | nsec | > 500 msec | | 31-60<br>Increa | | >60 m<br>Increa | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Treatment | Time | n | % | n r | | n % | Ś | n | % | n | % |
| QT interval | Treatment 1 | 1h | | | | | | | | | | |
| | (N=xx) | 2h | | | | | | | | | | |
| | | 3h | | | | | | | | | | |
| | Treatment 2 | 1h | | | | | | | | | | |
| | (N=xx) | 2h | | | | | | | | | | |
| | | 3h | | | | | | | | | | |
| QTcB interval | Treatment 1 | 1h | | | | | | | | | | |
| | (N=xx) | 2h | | | | | | | | | | |
| | | 3h | | | | | | | | | | |
| | Treatment 2 | 1h | | | | | | | | | | |
| | (N=xx) | 2h | | | | | | | | | | |
| | | 3h | | | | | | | | | | |

Source: Listing 16.2.xx

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all treatments, variables and time points.

#### Template T\_PE1

Table 14.3.8.xx Summary of Physical Examination Data

| | Planned | | | |
|--------------------|----------|--------------|-------------|-------------|
| | Relative | | Treatment 1 | Treatment 2 |
| Body System | Time | Result | (N=xx) | (N=xx) |
| General Appearance | Time 1 | Normal | n (%) | |
| | | Abnormal NCS | x (xx) | |
| | | Abnormal CS | | |
| | Time 2 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |
| HEENT | Time 1 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |
| | Time 2 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |

Source: Listing 16.2.xx

Programming notes: Continued with all body system, treatments and time points. Include rows for each outcome in CRF

If results are missing "missing" row will be added. Percentages calculated using the number of available results as denominator.

Template T\_NE1

Table 14.3.8.xx Summary of Neurological Examination Data

Mental Status

| | Planned | | | |
|-------------|----------|--------------|-------------|-------------|
| | Relative | | Treatment 1 | Treatment 2 |
| Body System | Time | Result | (N=xx) | (N=xx) |
| | | | n (%) | n (%) |
| Alertness | Time 1 | Normal | x (xx) | |
| | | Abnormal NCS | x (xx) | |
| | | Abnormal CS | | |
| | Time 2 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |
| Speech | Time 1 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |
| | Time 2 | Normal | | |
| | | Abnormal NCS | | |
| | | Abnormal CS | | |

Source: Listing 16.2.xx

Programming notes: Continued with all examinations/test, treatments and time points. Include rows for each outcome in CRF

For Ophthalmological assessment, replace body system with Test

If results are missing "missing" row will be added. Percentages calculated using the number of available results as denominator.

 ${\it Use PESCAT as subheading (not for Ophthalmological Assessment)}.$ 

Sponsor code: DNDI-EMO-001 Part 2

#### Template T\_PK1

Table 14..2.xx Summary of Emodepside Plasma Pharmacokinetic Concentration-Time Data [units]

| | | Planned<br>Relative | | No. | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Ν | Time | n | Imputed | Mean | 95% CI | SD | %CV | Median | Min | Max |
| Dose 1 | | 1h | | | | | | | | | |
| Oose 2 | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and timepoints

Means, SD, CI and CV should only be calculated if ≥2/3 individual values are >LLOQ

#### Template T\_PK3

Table 14..2.xx Summary of Derived Emodepside Plasma Pharmacokinetic Parameters

| _ | | | | 3-11-2 | 0.5 | 2/2/ | | | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter | Treatment | N n | Mean | 95% CI | SD | %CV | Median | Min | Max |
| AUC <sub>last</sub> (units) | | | | | | | | | |
| C <sub>max</sub> (units) | | | | | | | | | |
| max v | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and parameters

Sponsor code: DNDI-EMO-001 Part 2

Template T\_PK4

Table 14..2.xx Summary of Log-Transformed Derived Emodepside Plasma Pharmacokinetic Parameters

| Parameter | Treatment | N | n | Geom Mean | 95% CI | SD (logs) {%CVb} |
|---|---|---|---|---|---|---|
| AUC <sub>last</sub> (units)<br>C <sub>max</sub> (units) | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and parameters

Template T\_PK7

Table 14.2.xx Assessment of the Effects of Food on the PK of Emodepside

| Parameter | Treatment | Fed | Fasted | Ratio | 90% CI |
|---|---|---|---|---|---|
| | | | | Natio | 30/0 CI |
| | | | | (Fed/Fasted) | |
| Cmax (Units) | | xxxx.xx | XXXX.XX | xxxx.xx | (xxxx.xx, xxxx.xx) |

Source: Listing 16.2.xx

Programming notes: Continued with AUC<sub>inf</sub>,

#### Template T\_PD1

Table 14...xx Summary of Glucose

| | | | | | | | | | | Ch | ange f | rom Baselin | e | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | | | | | | | | | | | | | |
| Treatment | Relative Time | n | Mean | 95% CI | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Treatment 1 (N=xx) | -24h | х | x | x | х | x | х | х | | | | | | |
| | -20h | х | x | х | х | х | х | x | x | х | x | x | Х | х |

Note: Baseline on Day -1 is -24h value, baseline on Day 0 is Day 0, pre-dose

Programming notes: Continued with all PD parameters, treatments and timepoints

Change from baseline calculated from "pre-dose" on each day

### Template T\_PD2

Table 14...xx Summary of Difference Between Day -1 and Day 0 in Glucose

| | Planned Relative Time | | Day | -1 – Day | 0 |
|--------------------|-----------------------|---|------|----------|--------|
| Treatment | | n | Mean | SD | 95% CI |
| Treatment 1 (N=xx) | | | | | |

Note: Difference is change from baseline

Programming notes: Continued with time points and treatments

Sponsor code: DNDI-EMO-001 Part 2

## Template T\_PD3

Table 14...xx Summary of AUC<sub>0-24</sub> for change from baseline in Glucose (units)

| | Day -1 | | | | | Day 0 | | | | | Day -1 – Day 0 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | Mean | SD | Min | Max | n | Mean | SD | Min | Max | n | Mean | SD | 95% CI |
| Treatment 1 (N=xx) | | | | | | | | | | | | | | |

Note: Difference is change from baseline

Programming notes: Continued with all treatments

## 17.2.2 Figure Outlines

#### Template F\_PK1

Figure 16.2.4 .xx Individual Emodepside Plasma Concentration-Time Plots (Linear and Semi-log)



Programming note: Plot will include all subjects for a given treatment group

#### Template F\_PK2

Figure 16.2.4.xx Geometric mean (+ SD) of Emodepside Plasma Concentration-Time Plots (Linear and Semi-log)





Programming note: The SD is the geometric standard deviations

#### Template F\_PK10

Figure 16.2.xx Individual Emodepside Plasma Concentration-Time Plots (log scale) for Estimation of Lambda-z, with Regression Line



#### Template F\_PD1

Figure **16.2.**xx Individual Glucose-Time Plots



Programming note: Continue with Insulin, Glucagon and Cortisol land normal rages as reference lines.

For Blood pressure and Heart Rate, include PCI limits as reference lines.

Plot will include all subjects for a given treatment group

4 plots per page

### Template F\_PD2

Figure 16.2.xx Individual Glucose and PK Concentration Plots - Including Related Significantly Important AE Durations



Cohorts with at least 1 related significant AE displayed

Programming note: Continue with Insulin
2 plots per page

Sponsor code: DNDI-EMO-001 Part 2

## 17.2.3 Listing Outlines

#### Template L\_SD1\_PG

Listing 16.2.x.xx Listing of Study Dates

Treatment Subject Screening Day -1 Day 0 Follow-Up

Programming notes: Lists dates for screening, each dosing period and follow up

#### Template L\_SD2\_PG

Listing 16.2.x.xx Listing of Reasons for Withdrawal

Date of Study

Treatment Subject Withdrawal Day Reason

#### Template L\_DV1\_PG

Listing 16.2.x.xx Listing of Subjects with Inclusion/Exclusion Criteria Deviations

Treatment Subject Type Criterion
Inclusion

Exclusion

Hammersmith Medicines Research

Sponsor code: DNDI-EMO-001 Part 2

Template L\_TD1\_PG

Listing 16.2.x.xx Listing of Subjects with Time Deviations

Allowed Actual deviation deviation

Treatment Subject Timepoint Procedure (h:min) (h:min)

Programming notes: Only include time deviations which exceed the allowed deviation

Template L\_DV2\_PG

Listing 16.2.2.3 Listing of Subjects with Other Protocol Deviations

Treatment Subject Protocol Deviation

Template L\_AN1\_PG

Listing 16.2.x.xx Listing of Analysis Populations

Treatment Subject Safety Population PK concentration

Programming notes: continue for all populations

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_DM1\_PG

Listing 16.2.x.xx Listing of Demographic Characteristics

| | | | | | | | | | | | Alcohol | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Height | Weight | | Consumption | Cigarettes |
| Treatment | Subject | Date of visit | Date of birth | Age (y) | Gender | Race | Ethnicity | (cm) | (kg) | BMI (kg/m2) | (units/week) | (daily) |
| Treatment 1 | | | | | | | | | | | | |

. . . .

### Template L\_CM1\_PG

Listing 16.2.x.xx Listing of Concomitant Medications

| | | | Dose/ | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Drug Name/ | Units/ Freq/ | Date/time Started/ | Time Since Last | Started | Pre- | Ongoing |
| Treatment | Subject | Indication | Route | Date Stopped | Dose | Trial? | | Medication? |

#### Template L\_EX1\_PG

Listing 16.2.x.xx Listing of Exposure Data

| | | | | Dur- | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Start Date/ | Stop Date/ | ation | | Dose | Formulation | n/ |
| Treatment | Subject | Start Time of Dose | Stop Time of Dose | (days) | Dose | Unit | Route | Frequency |
| Treatment 1 | 1001 | 01JAN2002/ | 15FEB2002/ | 46 | 25 | mg | Tablet/ | 2xday |
| | | 23:59 | 15:30 | | | | Oral | |

## Template L\_AE1\_PG

Listing 16.2.x.xx Listing of All Adverse Events

| | | | | | | Frequency/ Action | Related to Study |
|---|---|---|---|---|---|---|---|
| | | SYSTEM ORGAN CLASS/ | Outcome/ Onset | | Severity/ | Taken (1)/ | Drug/ |
| | | PREFERRED TERM/ | Date/Time/ Resolved | Time Since Last | Serious/ | Other Action | Treatment |
| Treatment | Subject | Verbatim Text | Date/Time/ Duration | Dose | Withdrawal | Taken | Emergent? |
| Treatment 1 | 1001 | GASTROINTESTINAL | Resolved/ | 10d 7h 3m | Mild/ | Intermittent/ Dose | Possibly/ |
| | | DISORDERS / | 24SEP2003/13:05/ | | No/ | not changed/ | Yes |
| | | INTESTINAL SPASM/ | 27OCT2003/7:50/ | | Yes | None | |
| | | Entero-spasm | 34d 4h 5m | | | | |

<sup>(1)</sup> Action Taken with Study Treatment

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_LB1\_PG

Listing 16.2.x.xx Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance

| | | | Planned<br>Relative | | Study | | | | | Clinically |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Laboratory test (units) | Time | Date/Time | Day | Value | Normal Range | NR | BL | Significant? |
| Treatment 1 | 1001 | Alk Phos (U/L) | Time 1 | 01JAN2002/ | -1 | 64.00 | 32.0- 92.0 | | | |
| | | | | 13:34 | | | | | | |
| | | | Time 2 | 01APR2002/ | 85 | 84.00 | 32.0- 92.0 | | | |
| | | | | 07:22 | | | | | | |
| | | ALT (U/L) | Time 1 | 01JAN2002/ | -1 | 29.00 | 10.0- 40.0 | | | |
| | | | | 18:56 | | | | | | |
| | | | Time 2 | 01APR2002/ | 85 | 70.00 | 10.0- 40.0 | Н | - 1 | Υ |
| | | | | 09:22 | | | | | | |

NR for Normal Range flag, BL for Change from Baseline flag;

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Programming notes: Lists only double-flagged subjects

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_LB2\_PG

Listing 16.2.x.xx Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities

| | | Planned<br>Relative | | Alkaline | Phosphata | se (IU/L) | Alanine | Amino Tra<br>(IU/L) | nsferase | Aspartate | Amino Tran<br>(IU/L) | sferase | Total B | ilirubin (UN | MOL/L) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Time | Date/Time | Result | NR | BL | Result | NR | BL | Result | NR | BL | Result | NR . | BL |
| | | Planned | | | | | | | | | | | | | |
| | | Relative | | Chlo | ride (MMC | DL/L) | Gluc | ose (MMC | L/L) | Potas | sium (MMOL | L/L) | Sod | ium (MMO | L/L) |
| Treatment | Subject | Time | Date/Time | Result | NR | BL | Result | NR | BL | Result | NR | BL | Result | NR | BL |
| | | | Planned | | | | | | | | | | | | |
| | | | Relative | | | Calcium | (MMOL/L) | | Creatinin | e (UMOL/L) | | | Etc. | | |

NR for Normal Range flag, BL for Change from Baseline flag;

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Programming notes: Lists only double-flagged subjects

*Include all parameters for the study following the order from the lab report (above is a guide only)* 

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_URI

Listing 16.2.x.xx Listing of Urinalysis Data

| | | Planned | | Specific | Gravity | рН | 1 | Prot | ein | Glu | cose |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Relative | | | | | | | | | |
| Treatment | Subject | Time | Date/Time | Result | NR | Result | NR | Result | NR | Result | NR |

NR for Reference interval flag, H = Above reference interval, L = Below reference interval

Programming notes: Include all parameters for the study following the order from the lab report (above is a guide only)

#### Template L\_VS1\_PG

Listing 16.2.x.xx Listing of Vital Signs of Potential Clinical Importance

| | | | | Systolic | Diastolic | |
|---|---|---|---|---|---|---|
| | | Planned Relative | | Blood Pressure | Blood Pressure | Etc |
| Treatment | Subject | Time | Date/Time | (mmHg) | (mmHg) | (units) |
| | | 24 H | 26SEP2012:09:57 | 63 | 148* | |

<sup>\*</sup> Value of potential clinical importance

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_EG1\_PG

Listing 16.2.x.xx Listing of ECG Values of Potential Clinical Importance

| | | | | | | | QT Int | . (msec) | QTcB | (msec) | QTcF | (msec) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Subject | Planned<br>Relative Time | Date/Time | Heart<br>Rate<br>(bpm) | PR Int.<br>(msec) | QRS<br>Dur.<br>(msec) | QRS<br>Axis<br>(deg) | Observed | Change<br>from<br>Baseline | Observed | Change<br>from<br>Baseline | Observed | Change<br>from<br>Baseline |
| | Pre-dose (1) | 26SEP2012:09:57 | 63 | 148 | 78 | 50 | 390 | 32.7 * | 399 | -27.7 | 419 | -11 |
| | Pre-dose (2) | | | | | | | | | | | |
| | Pre-dose (3) | | | | | | | | | | | |
| | Mean Pre-dose | | | | | | | | | | | |
| | 24 H | | | | | | | | | | | |

<sup>\*</sup> Value of potential clinical importance

Programming notes: Do not list RR

#### Template L\_EG2\_PG

Listing 16.2.x.xx Listing of Abnormal ECG Findings

| | | | | | Comment on |
|---|---|---|---|---|---|
| | | Planned Relative | | | Clinical |
| Treatment | Subject | Time | Date/Time | ECG Finding | Significance |

Programming notes: Lists only values with Normal variant='No' or with comment on ECG result

ECG Finding contains Physician's Opinion from CRF and relates to whole trace (not individual parameters), e.g. Normal, Abnormal - NCS or Abnormal - CS

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_PE1\_PG

Listing 16.2.x.xx Listing of Abnormal Physical Examination Findings

Planned Relative

Treatment Subject Time Date/Time Site Details

Programming Notes: List only findings with an 'Abnormal NCS' or 'Abnormal CS' result.

If subjects have multiple abnormal sites at a given time, create a separate row for each site.

#### Template L\_NE1\_PG

Listing 16.2.x.xx Listing of Neurological Examination Findings

Planned

Treatment Subject Relative Time Date/Time Type Assessment Details

Programming Notes: Type = (Mental Status, Mood, Cranial Nerves etc.

List all findings

If subjects have multiple abnormal assessment at a given time, create a separate row for each assessment.

For Ophthalmological assessment, the columns will be Treatment, Subject, Planned relative Time, Date/Time, Test and Details

#### Template L\_NE2\_PG

Listing 16.2.x.xx Listing of Neurological Questionnaire Findings

Mental Status

Total Score
Hamilton Epworth

Planned Relative Depression Sleepiness

Treatment Subject Time Date/Time Rating Scale Score BDI-II

Sponsor code: DNDI-EMO-001 Part 2

#### Template L\_PK1\_PG

Treatment

Listing 16.2.4.xx Listing of Emodepside Plasma Pharmacokinetic Con centration-Time Data

{Add.

time Planned var.} Date Study Day Relative Time

Time Deviation Actual Relative (units) Time

Time Concentration (units)

BLQ = Below Limit of Quantification

Actual time

Programming notes: Values below LLOQ are shown as BLQ

Subject

For PD: BLQ values are imputed to half LLOQ

For the listings of derived AUCO-24 PD concentrations, the columns will be Treatment, Subject, Planned Relative Time, Concentrations (units)

#### Template L\_PK3\_PG

Listing 16.2.4 xx Listing of Emodepside Urine Excretion Rate Data

Planned

Relative

Urine Conc.

Treatment Subject Time Start Date/Time Stop Date/Time (units) Total Sample Volume (mL) Amount excreted (units)

#### Template L\_PK4\_PG

Listing 16.2.4.xx Listing of Derived Emodepside Pharmacokinetic Parameters

{Add.

Programming notes: Continue with all parameters

# **Appendix A: Laboratory Ranges**

# Pre-determined Changes for Laboratory Data (from FL140 v3)

| | | | | Delta ranges | |
|---|---|---|---|---|---|
| Test | Test Code | Unit | Sex | Acceptable | Acceptable |
| | 1 cst couc | | SCA | decrease | increase |
| Activated partial thromboplastin time | APTTT | sec | Both | - 8.0 | + 8.0 |
| Alanine transferase | ALTN | IU/L | F | - | + 30 |
| Alanine transferase | ALTN | IU/L | M | - | + 30 |
| Albumin | ALB | g/L | Both | - 7.5 | + 7.5 |
| Alkaline phosphatase | ALPN | IU/L | Both | - 30 | + 30 |
| Amylase | AMY | U/L | Both | - | + 150 |
| Aspartate transferase | ASTN | IU/L | F | - 30 | + 30 |
| Aspartate transferase | ASTN | IU/L | M | - 30 | + 30 |
| Basophils | BASO | 10 <sup>9</sup> /L | Both | - | + 0.3 |
| Bilirubin conjugated | DBIL | μmol/L | Both | - | + 4.0 |
| Bilirubin total | TBIL | μmol/L | F | - 20 | + 10.0 |
| Bilirubin total | TBIL | μmol/L | M | - 20 | + 10.0 |
| Bilirubin unconjugated | IBIL | μmol/L | Both | - | - |
| C-reactive protein | CRP | mg/L | Both | - | - |
| CK relative index | CKMBR | % | Both | - | - |
| Calcium | CA | mmol/L | Both | - 0.4 | + 0.4 |
| Carbon dioxide | CO2 | mmol/L | Both | - 8 | + 8 |
| Chloride | CL | mmol/L | Both | - 10 | + 10 |
| Cholesterol | CHOL | mmol/L | Both | - | + 0.7 |
| Creatine kinase | CK | IU/L | F | - | + 400 |
| Creatine kinase | CK | IU/L | M | - | + 400 |
| Creatinine | CREA | μmol/L | Both | - | + 40 |
| Creatinine (DOA urine) | CREDA-U | mmol/L | Both | - | - |
| Eosinophils | EOS | 10 <sup>9</sup> /L | Both | - | + 0.5 |
| Erythrocyte sedimentation rate | ESR | mm/h | Both | - | - |
| Fibrinogen | FIB-C | g/L | Both | - | - |
| Free T3 | FT3 | pmol/L | Both | - 3.5 | + 3.5 |
| Free T4 | FT4 | pmol/L | Both | - 15 | + 15 |
| Gamma glutamyl transferase | GGT | IU/L | F | - | + 40 |
| Gamma glutamyl transferase | GGT | IU/L | M | - | + 40 |
| Globulin | GLOB | g/L | Both | - 7.5 | - |
| Glucose | GLU | mmol/L | Both | - 1.5 | + 2.5 |
| Haematocrit | HCT | L/L | Both | - 0.05 | - |
| Haemoglobin | HB | g/L | Both | - 20 | - |
| High density lipoprotein | HDL | mmol/L | Both | - 1.5 | + 1.5 |
| International normalised ratio | INRR | ratio | Both | - | - |
| Lactate dehydrogenase | LDH | IU/L | Both | - | + 150 |
| Lymphocytes | LYMP | 10 <sup>9</sup> /L | Both | - 1.5 | + 1.5 |
| Magnesium | MG | mmol/L | Both | - | - |
| Mean cell haemoglobin | MCH | pg | Both | - 2 | + 2 |
| Mean cell haemoglobin concentration | MCHC | g/L | Both | - 25 | + 25 |
| Mean cell volume | MCV | fL | Both | - 10 | + 10 |
| | | | 1 | | 1 |

| | | | | Delta | ranges |
|---|---|---|---|---|---|
| Test | Test Code | Unit | Sex | Acceptable decrease | Acceptable increase |
| Monocytes | MONO | 10 <sup>9</sup> /L | Both | - 0.50 | + 0.5 |
| Neutrophils | NEUT | 10 <sup>9</sup> /L | Both | - 2 | + 8 |
| Phosphate | PHOS | mmol/L | Both | - 1 | + 1 |
| Platelets | PLT | 10 <sup>9</sup> /L | Both | - 100 | + 100 |
| Platelets (citrate tube) | PLTC | 10 <sup>9</sup> /L | Both | - 100 | + 100 |
| Potassium | K | mmol/L | Both | - 0.75 | + 0.75 |
| Prolactin | PROL | μg/L | Both | - | - |
| Prothrombin time | PTT | sec | Both | -4.0 | + 4.0 |
| Red blood cells | RBC | $10^{12}/L$ | Both | - 1.0 | - |
| Reticulocyte | RET | % | Both | - | - |
| Reticulocyte count | RETC | 10 <sup>9</sup> /L | Both | - | - |
| Reticulocyte manual count | RETM | 10 <sup>9</sup> /L | Both | - | - |
| Sodium | NA | mmol/L | Both | - 8 | + 8 |
| Thrombin time | TT | sec | Both | - | - |
| Thyroid stimulating hormone | TSH | mIU/L | Both | - 3 | + 3 |
| Total protein | TP | g/L | Both | - 15 | - |
| Triglycerides | TG | mmol/L | Both | - | + 1.5 |
| Urea | UREA | mmol/L | Both | - 5 | + 2 |
| Uric acid | UA | μmol/L | Both | - 100 | + 100 |
| Urine pH | UPH | N/A | Both | -4 | + 4 |
| Urine red blood cells | URBC | $10^{6}/L$ | Both | - | + 10 |
| Urine white blood cells | UWBC | $10^{6}/L$ | Both | - | + 100 |
| White blood cells | WBC | 10 <sup>9</sup> /L | Both | - 2 | + 8 |

## **Appendix B: Pharmacokinetic Analysis**

## 1 Calculation Methods

# 1.1 Data Handling Conventions

#### 1.1.1 Actual v Planned Times

Actual sample times will be used for the calculation of pharmacokinetic parameters and for individual concentration-time plots.

Planned sampling times will be used to calculate the concentration-time summary statistics and summary concentration-time plots.

### 1.1.2 Missing and BQL Concentrations

Missing values will not be used in any way.

For calculation of all pharmacokinetic parameters and individual profile plots, plasma concentrations below the quantifiable limit (BQL) of the assay will not be used for the calculation of PK parameters (except BQL values observed at time points before the maximum concentration, which will be taken as zero).

BQL values will be substituted by one half of the lower limit of quantification for calculation of plasma concentration summary statistics. The number of imputed values will be included in the summary table.

For urine concentrations reported as BQL it is not possible to impute a value. The amount excreted will be set to zero when concentration is BQL.

#### 1.2 AUC Calculations

The AUC will be calculated by a combination of linear and logarithmic methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations

 $AUC_{(0-\infty)}$  values with <20% of this area extrapolated will be reported.

It is acceptable to include data from profiles with >20% extrapolated as long as at least 80% of the profiles in the study have <20% of the  $AUC_{(0-\infty)}$  as extrapolated area. In this instance, individual plasma concentration-time profiles for which the extrapolated

It is unacceptable to use  $AUC_{(0-\infty)}$  data if >40% of the AUC has been extrapolated, except in specific situations which should be carefully justified in the study report.

#### 1.3 Lambda-z Calculations

areas are >20% of AUC<sub>(0- $\infty$ )</sub> will be identified.

The apparent terminal phase rate-constant ( $\lambda_z$ ) will be estimated by linear regression of logarithmically transformed concentration versus time data. Only those data points which are judged to describe the terminal log-linear decline will be used in the regression.

During the analysis, repeated regressions are carried out using the last three points with non-zero concentrations, then the last four points, last five, etc. Points prior to  $C_{max}$  are not used. Points with a value of zero for the concentration are excluded. For each regression, an adjusted  $R^2$  is computed. The  $\lambda_z$  using the regression with the largest adjusted  $R^2$  is selected. If the adjusted  $R^2$  does not improve, but is within 0.0001 of the largest adjusted  $R^2$  value, the regression with the larger number of points is used.  $\lambda_z$  must be positive, and calculated from at least three data points.

For non-compartmental analysis uniform weighting will be applied.

#### 1.4 Observed v Predicted Values

For parameters dependent on  $\lambda_z$ , the 'predicted' rather than the 'observed' parameters will be calculated.

The 'predicted' parameters are calculated using  $\hat{C}_t$  (the predicted value of the concentration at time tn); whilst the 'observed' parameters use the last observed concentration.

# 2 General Considerations for Data Analysis

### 2.1 Derived and transformed data

In general, concentration and concentration-related quantities, rate constants and half-lives (e.g.  $C_{max}$ , AUC,  $t_{1/2}$ , CL/F,  $V_z$ /F and MRT) will be analysed after logarithmic transformation. Logarithmic transformations will use natural logarithms (log<sub>e</sub>). A list of those parameters that will be log transformed are given below.

## 2.2 Summary data

Means at any time will only be calculated if at least 2/3 of the individual data are measured and are above the lower of quantification (LLOQ).

# 3 Parameter Definitions

## 3.1 Plasma Parameters

# 3.1.1 Emodepside

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| Concentrations and | | | | | | | |
| C <sub>max</sub> | Maximum (peak) plasma concentration | The maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | ng/mL | Y | Cmax | CMAX | $\mathrm{C}_{\mathrm{max}}$ |
| C <sub>max</sub> /D | Dose-normalised C <sub>max</sub> to infinity | The dose-normalised $C_{max}$ will be calculated as $C_{max}$ /Dose administered | (ng/mL)/mg | Y | Cmax_D | CMAXD | C <sub>max</sub> /D |
| $C_{max,norm}$ | Observed maximum plasma concentration corrected by dose and body weight | The C <sub>max</sub> normalised by dose and body weight will be calculated as C <sub>max</sub> /(Dose administered*body weight) | (ng/mL)/(mg*kg) | Y | N/A | CMAXWD | $C_{	ext{max,norm}}$ |
| t <sub>max</sub> | Time to reach maximum (peak) plasma concentration | The first time of maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | h | N | Tmax | TMAX | t <sub>max</sub> |
| Half-life | | | | | | | |
| $\lambda_z$ | Terminal rate constant | The apparent terminal phase rate-constant $(\lambda_z)$ will be estimated by linear regression of logarithmically transformed concentration versus time data. | 1/h | Y | Lambda_z | LAMZ | $\lambda_{\mathrm{z}}$ |
| Point terminal | Number of points for<br>Lambda z | The number of time points used in calculating Lambda z | - | - | No_points_lambda<br>_z | LAMZNPT | $n_{pts}$ |
| t <sub>1/2</sub> | Terminal half-life | The terminal half-life calculated from the terminal slope of the log concentration-time curve, as follows: $t_{1/2} = \frac{\log_e 2}{\lambda_z}$ | h | Y | HL_Lambda_z | LAMZHL | t <sub>1/2</sub> |
| t <sub>½,0-24</sub> | Dominant half-life | The half-life calculated from the terminal slope of the log concentration-time (0-24h) curve, as follows: $t_{1/2} = \frac{\log_e 2}{\lambda_z}$ | h | Y | HL_Lambda_z | TBC | t <sub>1/2,0-24</sub> |

Sponsor code: DNDI-EMO-001 Part 2

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| Areas under the cur | . , . | | | | | | |
| AUCt | Area under the plasma concentration-time curve from time zero to time of last measurable concentration | The area under the concentration-time curve from zero time (pre-dose) to the time of last quantifiable concentration will be calculated using the (specified) trapezoidal method. | h*ng/mL | Y | AUClast | AUCLST | AUC <sub>last</sub> |
| $\mathrm{AUC}_{\mathrm{t,norm}}$ | Area under the concentration-time curve from time zero (pre-dose) to the time of last quantifiable concentration corrected by dose and body weight | The AUC normalised by dose and body weight will be calculated as AUC <sub>t</sub> /(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | N/A | AUCLSTWD | AUC <sub>last,norm</sub> |
| AUC <sub>1-∞</sub> | Area under the exponential curve from t <sub>last</sub> to infinity | The area under the exponential curve from $t_{last}$ to infinity, calculated as follows: $AUC_{t-\infty} = \frac{\hat{C}_t}{\lambda_z} \text{ where } \hat{C}_t \text{ is the }$ predicted value of the concentration at $t_{last}$ . | h*ng/mL | N/A | N/A | AUCIFO | AUCt-inf |
| $\mathrm{AUC}_{\infty}$ | Area under the plasma concentration-time curve from time zero to infinity | The area under the concentration-time curve will be calculated using the (specified) trapezoidal method for the interval 0 to t <sub>last</sub> (time t <sub>last</sub> is the time at which the last non-zero level was recorded), plus AUC <sub>1-∞</sub> . | h*ng/mL | Y | AUCINF_pred | AUCIFP | AUC <sub>inf</sub> |
| AUC∞/Dose | Dose-normalised AUC to infinity | The dose-normalised AUC to infinity will be calculated as AUC <sub>∞</sub> /Dose administered | (h*ng/mL)/mg | Y | AUCINF_D_pred | AUCIFPD | AUC <sub>inf</sub> /D |
| $\mathrm{AUC}_{\infty,\mathrm{norm}}$ | Area under the concentration-time curve from time zero to infinity corrected by dose and body weight | The AUC normalised by dose and body weight will be calculated as AUC <sub>x</sub> /(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | N/A | AUCIFPWD | AUC <sub>inf,norm</sub> |
| %AUC <sub>extrap</sub> | Percentage of $AUC_{\infty}$ extrapolated from from $t_{last}$ to infinity | $\% AUC_{extrap} = \frac{100 \times AUC_{t-\infty}}{AUC_{\infty}}$ | % | N | AUC_%EXTRAP<br>_pred | AUCPEP | %AUC <sub>extrap</sub> |

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| AUC <sub>0-24</sub> | Area under the plasma concentration-time curve from time zero to 24h | The area under the concentration-time curve from zero time (pre-dose) to 24h will be calculated using the (specified) trapezoidal method. If $\lambda_z$ is not estimable, a partial AUC is not calculated (when $t_{last} < t$ ). | h*ng/mL | Y | User specified area | AUCINT | AUC <sub>24</sub> |
| AUC <sub>0-24</sub> /D | Dose-normalised AUC from time zero to 24h | The dose-normalised AUC from time zero to 24h will be calculated as AUC <sub>0-24</sub> /Dose administered | (h*ng/mL)/mg | Y | N/A | AUCINTD | AUC <sub>24</sub> /D |
| AUC <sub>0-24,norm</sub> | Area under the concentration-time curve from time zero to 24h corrected by dose and body weight | The AUC from time zero to 24h normalised by dose and body weight will be calculated as AUC <sub>0-24</sub> /(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | N/A | AUCINTWD | AUClast,norm |
| | f distribution and mean residen | | | | | | |
| CL/F | Apparent total clearance from plasma after oral administration | Apparent total clearance from plasma will be calculated using the following formula: $CL/F = \frac{Dose}{AUC_{\infty}}$ | L/h | Y | Cl_pred (actually derives Cl_F_pred for oral dose) | CLFP | CL/F |
| V <sub>z</sub> /F | Apparent volume of distribution during terminal phase after non-intravenous administration | Apparent volume of distribution will be calculated using the following formula: $V_z / F = \frac{Dose}{\lambda_z \bullet AUC_{\infty}}$ | L | Y | Vz_pred (actually derives Vz_F_pred for oral dose) | VZFP | V <sub>z</sub> /F |
| MRT | Mean Residence Time | The mean residence time will be calculated using: $MRT = \frac{AUMC}{AUC_{\infty}}$ | h | Y | MRTINF_pred | MRTIFP | MRT |
| AUMC | Area under the first moment of the plasma concentration-time curve from time zero to infinity | The area under the first moment of the concentration-time curve from zero time (predose) extrapolated to infinite time will using the (specified) trapezoidal method, as for AUC. | h <sup>2</sup> *ng/mL | - | AUMCINF_pred | AUMCIFP | AUMC |

Sponsor code: DNDI-EMO-001 Part 2

# **Appendix C: Sample Page Layout**

| DNDi: DNDI-EMO-001 | | Page x of y* |
|---|---|---|
| Population: [Pop] | | |
| | Table [number] [title] | |
| | Column headers | |
| | Main body of output | |
| | Source: Listing [16.2.xx] | |
| Footnotes about the table or listing text go here. | | |
| Program: [Prog Name] Produced By:[Username] | [Date] | HMR 15-020 Part 2 |

Font size will be Arial 9.5pt. The following margins will be used: Left: 1", Right: 1", Top: 1", Bottom: 1"

<sup>\*</sup>y = last page of individual output